CLINICAL TRIAL: NCT01643928
Title: EXTENSION STUDY EVALUATING TREATMENT WITH PF-05280586 VERSUS RITUXIMAB IN SUBJECTS WITH ACTIVE RHEUMATOID ARTHRITIS WHO HAVE PARTICIPATED IN OTHER PF-05280586 CLINICAL TRIALS
Brief Title: Rheumatoid Arthritis Extension Trial For Subjects Who Have Participated In Other PF-05280586 Trials (REFLECTIONS B328-04)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Masking: Triple | Purpose: Treatment
Other Study IDs: B3281004; ICON 9002/0101; 2012-003223-38 (EudraCT Number)
Record Dates: First submitted 2012-07-06; First posted 2012-07-18 (Estimated); Results first posted 2017-06-08 (Actual); Last update posted 2019-01-29 (Actual); Status verified 2019-01

CONDITIONS: Rheumatoid Arthritis
Keywords: extension trial; rheumatoid arthritis; rituximab
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Rituximab-Pfizer (Experimental)
  Interventions: Biological: Rituximab-Pfizer (PF-05280586) x 3 courses
- Rituximab-EU+Rituximab-Pfizer (Active Comparator): Subjects will receive Rituximab-EU x 1 course followed by Rituximab-Pfizer x 2 courses.
  Interventions: Biological: Rituximab-EU+ Rituximab-Pfizer x 2 Courses
- Rituximab-US+Rituximab-Pfizer (Active Comparator): Subjects will receive Rituximab-US x 1 course followed by Rituximab-Pfizer x 2 courses.
  Interventions: Biological: Rituximab-US + Rituximab-Pfizer x 2 Courses

INTERVENTIONS:
Biological: Rituximab-Pfizer (PF-05280586) x 3 courses — 1000 mg intravenous infusion [IV] on Days 1 and 15 of each 24 week treatment course for up to 3 treatment courses
  Arms: Rituximab-Pfizer
Biological: Rituximab-EU+ Rituximab-Pfizer x 2 Courses — Subjects will receive Rituximab-EU x 1 course followed by Rituximab-Pfizer x 2 courses. 1000 mg IV infusion of Rituximab-EU on Days 1 and 15 of a 24 week treatment course followed by 1000 mg IV infusion of PF-05280586 on Days 1 and 15 of each 24 week course for up to 2 additional treatment courses
  Arms: Rituximab-EU+Rituximab-Pfizer
Biological: Rituximab-US + Rituximab-Pfizer x 2 Courses — Subjects will receive Rituximab-US x 1 course followed by Rituximab-Pfizer x 2 courses. 1000 mg IV infusion of Rituximab-US on Days 1 and 15 of a 24 week treatment course followed by 1000 mg IV infusion of PF-05280586 on Days 1 and 15 of each 24 week course for up to 2 additional treatment courses
  Arms: Rituximab-US+Rituximab-Pfizer

SUMMARY:
This extension study will evaluate the safety (including immunogenicity) of treatment with rituximab-Pfizer, as well as the safety and immunogenicity after transitioning from rituximab-US or rituximab-EU to rituximab-Pfizer. This study will provide continued treatment access to subjects with active rheumatoid arthritis who have participated for at least 16 weeks in other studies in the rituximab Pfizer program.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.
* Participated for a minimum of 16 weeks after the initiation of the last course of treatment in a previous rheumatoid arthritis study in the rituximab-Pfizer program within the past 2 months.

Exclusion Criteria:

* Investigational site staff members or relatives of those site staff members or subjects who are Pfizer employees directly involved in the conduct of the study.
* Initiated treatment with investigational agents or other biologics (including Rituxan and MabThera) since participating in a previous rheumatoid arthritis study in the rituximab-Pfizer program.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2012-08-16 (Actual); Primary Completion 2016-03-14 (Actual); Study Completion 2016-03-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (71):
- United States (34):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Rheumatology Associates of North Alabama, PC, Huntsville, Alabama
  - Arthrocare, Arthritiscare & Research, PC, Gilbert, Arizona
  - CHI St. Vincent Medical Group Hot Springs, Hot Springs, Arkansas
  - UCLA Clinical & Translational Research Center, Los Angeles, California
  - UCLA David Geffen School of Medicine, Los Angeles, California
  - Desert Medical Advances, Palm Desert, California
  - New England Research Associates, LLC, Trumbull, Connecticut
  - QPS Labs, Newark, Delaware
  - University of South Florida - College of Medicine Carol and Frank Morsani Center, Tampa, Florida
  - Loyola University Medical Center, Maywood, Illinois
  - Illnois Bone & Joint Institute, Morton Grove, Illinois
  - Covance Central Laboratory Services, Indianapolis, Indiana
  - Bluegrass Community Research, Inc., Lexington, Kentucky
  - Klein & Associates, M.D., P.A., Cumberland, Maryland
  - Clinical Pharmacology Study Group, Worcester, Massachusetts
  - Bronson Internal Medicine and Rheumatology, Battle Creek, Michigan
  - Justus J. Fiechtner, MD, PC, Lansing, Michigan
  - University of Nevada School of Medicine, Las Vegas, Nevada
  - Dartmouth - Hitchcock Medical Center, Lebanon, New Hampshire
  - North Shore-LIJ Health System - Division of Rheumatology and Allergy-Clinical, Great Neck, New York
  - PMG Research of Hickory LLC, Hickory, North Carolina
  - PMG Research of Hickory, LLC, Hickory, North Carolina
  - Cincinnati Rheumatic Disease Study Group, Cincinnati, Ohio
  - Health Research of Oklahoma, Oklahoma City, Oklahoma
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - The Arthritis Group, Philadelphia, Pennsylvania
  - Clinical Research Center of Reading, LLC, Wyomissing, Pennsylvania
  - Arthritis Associates, PLLC, Hixson, Tennessee
  - Arthritis Clinic, Jackson, Tennessee
  - West Tennessee Research Institute, Jackson, Tennessee
  - Metroplex Clinical Research Center, Dallas, Texas
  - Apocell, Inc, Houston, Texas
  - Southwest Rheumatology Research, LLC, Mesquite, Texas
- Rheumatology Research Unit, Maroochydore, Queensland, Australia
- Canada (4):
  - Pharmacie Matte et Petit, Québec, Quebec
  - Centre de Recherche Saint-Louis, Québec, Quebec
  - Clinique Medicale du Phare (ECG Only), Rimouski, Quebec
  - Centre de Rhumatologie de l'Est du Quebec, Rimouski, Quebec
- Colombia (10):
  - Clínica Medellín S.A. Sede Centro, Medellín, Antioquia
  - IPS Rodrigo Botero S.A.S., Medellín, Antioquia
  - Mix Supplier S.A., Medellín, Antioquia
  - Rodrigo Botero S.A.S., Medellín, Antioquia
  - Centro de Reumatologia y Ortopedia, Barranquilla, Atlántico
  - Clinica de La Costa Ltda., Barranquilla, Atlántico
  - Congregación de las Hermanas Franciscanas Misioneras de María Auxiliadora-Clinica La Asuncion, Barranquilla, Atlántico
  - IPS Centro Integral de Reumatologia del Caribe, CIRCARIBE S.A.S., Barranquilla, Atlántico
  - IPS Centro Integral De Reumatologia del Caribe, CIRCARIBE S.A.S, Barranquilla, Atlántico
  - Organizacion Clinica General Del Norte S.A., Barranquilla, Atlántico
- Schlosspark-Klinik GmbH, Internal Medicine II, Berlin, Germany
- The Chaim Sheba Medical Center, Tel Litwinsky, Israel
- Mexico (7):
  - Hospital Bernardette (Emergencies), Guadalajara, Jalisco
  - Private Office, Guadalajara, Jalisco
  - C.T. Scanner de Mexico, S.A. de C.V. (CT ONLY), Mexico City, Mexico City
  - CLIDITER, S.A de C.V., Mexico City, Mexico City
  - Hospital Angeles Clinica Londres, Mexico City, Mexico City
  - Hospital Angeles, Centro Medico del Potosi, San Luis Potosí City
  - Centro de Alta Especialidad en Reumatologia e Investigacion del Potosi, S.C., San Luis Potosí City
- Russia (10):
  - LLC Scientific and Research Medical Complex "Your Health", Kazan', Tatarstan Republic
  - State Institution of Healthcare "Regional Clinical Hospital for Wars' Veterans", Kemerovo
  - LLC Consulting and Diagnostic Rheumatological Center "Healthy Joints", Novosibirsk
  - St. Petersburg State Healthcare Institution "Clinical Rheumatology Hospital 25", Saint Petersburg
  - "AVA-PETER" Ltd - Affiliate Address, Saint Petersburg
  - AVA-PETER Ltd., Saint Petersburg
  - Local Ethics Committee of LLC AVA-PETER, Saint Petersburg
  - Laboratory of LLC AVA-PETER, Saint Petersburg
  - State Budget Institution of Healthcare "Samara Regional Clinical Hospital named after V.D. Seredavin, Samara
  - State Institution of Healthcare "Samara Regional Clinical Hospital named after V.D. Seredavin", Samara
- South Africa (2):
  - Panorama Medical Centre - Room 136, Cape Town
  - Dr. Jan Fourie Medical Centre, KwaZulu Natal
- Division of Rheumatic & Musculoskeletal Diseases, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Cohen SB, Burgos-Vargas R, Emery P, Jin B, Cronenberger C, Vazquez-Abad MD. Extension Study of PF-05280586, a Potential Rituximab Biosimilar, Versus Rituximab in Subjects With Active Rheumatoid Arthritis. Arthritis Care Res (Hoboken). 2018 Nov;70(11):1598-1606. doi: 10.1002/acr.23586. PMID 29692005
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B3281004&StudyName=Rheumatoid%20Arthritis%20Extension%20Trial%20For%20%20Subjects%20Who%20Have%20Participated%20In%20Other%20PF-05280586%20Trials%20%28REFLECTIONS%20B328-04%29%20

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an extension study for participants with active rheumatoid arthritis who had participated for at least 16 weeks in a prior rituximab-Pfizer protocol (B3281001) and had not received intervening treatment with investigational agents or other biologics (including Rituxan and MabThera).
Pre-assignment Details: Participants given PF-05280586 in Study B3281001 received PF-05280586. Participants given licensed product in Study B3281001 received the same licensed product or PF-05280586 in Course 1. All participants received PF-05280586 in later courses. 185 participants were randomized to Study B3281004, 183 participants received study treatment.
Groups:
- PF-05280586/PF-05280586/PF-05280586: This group received intravenous (IV) rituximab (PF-05280586) infusion 1000 mg/500 mL (preceded by 100 mg IV methylprednisolone or its equivalent, an antipyretic, and an antihistamine) on Study Days 1 and 15 of up to 3 24-week (±8 week) courses. Participants continued to receive a stable background regimen of methotrexate 10 to 25 mg/week (7.5 mg/week in the event of prior poor tolerance). Folate supplementation was encouraged according to local standard of care. Participants in this treatment arm received PF-05280586 in the B3281001 study.
- Rituximab-EU/PF-05280586/PF-05280586: This group received IV rituximab (MabThera) infusion 1000 mg/500 mL (preceded by 100 mg IV methylprednisolone or its equivalent, an antipyretic, and an antihistamine) on Study Days 1 and 15 of a 24-week (±8 week) course followed by IV rituximab (PF-05280586) infusion 1000 mg/500 mL (preceded by 100 mg IV methylprednisolone or its equivalent, an antipyretic, and an antihistamine) on Study Days 1 and 15 of up to 2 24-week (±8 week) courses. Participants continued to receive a stable background regimen of methotrexate 10 to 25 mg/week (7.5 mg/week in the event of prior poor tolerance). Folate supplementation was encouraged according to local standard of care. Participants in this treatment arm received Rituximab-EU in the B3281001 study.
- PF-05280586/PF-05280586/PF-05280586 (EU): This group received IV rituximab (PF-05280586) infusion 1000 mg/500 mL (preceded by 100 mg IV methylprednisolone or its equivalent, an antipyretic, and an antihistamine) on Study Days 1 and 15 of up to 3 24--week (±8 week) courses. Participants continued to receive a stable background regimen of methotrexate 10 to 25 mg/week (7.5 mg/week in the event of prior poor tolerance). Folate supplementation was encouraged according to local standard of care. Participants in this treatment arm received Rituximab-EU in the B3281001 study.
- Rituximab-US/PF-05280586/PF-05280586: This group received IV rituximab (Rituxan) infusion 1000 mg/500 mL (preceded by 100 mg methylprednisolone, an antipyretic, and an antihistamine) on Study Days 1 and 15 of a 24--week (±8 week) course followed by IV rituximab (PF-05280586) infusion 1000 mg/500 mL (preceded by 100 mg IV methylprednisolone or its equivalent, an antipyretic, and an antihistamine) on Study Days 1 and 15 of up to 2 24-week (±8 week) courses. Participants continued to receive a stable background regimen of methotrexate 10 to 25 mg/week (7.5 mg/week in the event of prior poor tolerance) for up to 25 weeks. Folate supplementation was encouraged according to local standard of care. Participants in this treatment arm received Rituximab-US in the B3281001 study.
- PF-05280586/PF-05280586/PF-05280586 (US): This group received IV rituximab (PF-05280586) infusion 1000 mg/500 mL (preceded by 100 mg IV methylprednisolone or its equivalent, an antipyretic, and an antihistamine) on Study Days 1 and 15 of up to 3 24-week (±8 week) courses. Participants continued to receive a stable background regimen of methotrexate 10 to 25 mg/week (7.5 mg/week in the event of prior poor tolerance). Folate supplementation was encouraged according to local standard of care. Participants in this treatment arm received Rituximab-US in the B3281001 study.
Period: Overall Study
Arm/Group | PF-05280586/PF-05280586/PF-05280586 | Rituximab-EU/PF-05280586/PF-05280586 | PF-05280586/PF-05280586/PF-05280586 (EU) | Rituximab-US/PF-05280586/PF-05280586 | PF-05280586/PF-05280586/PF-05280586 (US)
Started | 58 | 32 | 33 | 30 | 30
Completed | 48 | 30 | 30 | 27 | 28
Not Completed | 10 | 2 | 3 | 3 | 2
Not completed — Lost to Follow-up | 1 | 0 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 1 | 0
Not completed — Pregnancy | 0 | 0 | 0 | 1 | 0
Not completed — Other | 5 | 1 | 1 | 0 | 0
Not completed — Adverse Event | 2 | 1 | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- PF-05280586/PF-05280586/PF-05280586: This group received IV rituximab (PF-05280586) infusion 1000 mg/500 mL (preceded by 100 mg IV methylprednisolone or its equivalent, an antipyretic, and an antihistamine) on Study Days 1 and 15 of up to 3 24-week (±8 week) courses. Participants continued to receive a stable background regimen of methotrexate 10 to 25 mg/week (7.5 mg/week in the event of prior poor tolerance). Folate supplementation was encouraged according to local standard of care. Participants in this treatment arm received PF-05280586 in the B3281001 study.
- Total: Total of all reporting groups
Arm/Group | PF-05280586/PF-05280586/PF-05280586 | Rituximab-EU/PF-05280586/PF-05280586 | PF-05280586/PF-05280586/PF-05280586 (EU) | Rituximab-US/PF-05280586/PF-05280586 | PF-05280586/PF-05280586/PF-05280586 (US) | Total
Number analyzed (Participants) | 58 | 32 | 33 | 30 | 30 | 183
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.3 (12.01) | 56.0 (11.88) | 56.7 (9.35) | 52.6 (13.73) | 55.8 (10.35) | 55.3 (11.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 29 | 23 | 20 | 25 | 147
  Male | 8 | 3 | 10 | 10 | 5 | 36

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants by Anti-Drug Antibody (ADA) Status Using Anti-PF-05280586 Antibody Assay
Description: Serum samples were collected to determine the presence of ADA using two validated assays, one specific for PF-05280586 and one specific for the licensed drug products. For participants assigned to PF-05280586 in Study B3281001, blood samples were screened for ADA using the assay specific to PF-05280586; if the blood samples were confirmed to be positive (+ve) for ADA against PF-05280586, the samples were also analyzed using the assay specific for the licensed drug products to assess cross-reactivity of the ADA. For participants assigned to the licensed products in Study B3281001, blood samples were screened for ADA using both assays in order to assess any product-specific ADA and/or cross-reactivity for the transition from the licensed products to PF-05280586.
Time Frame: Course 1 (C1) Overall, Course 2 (C2) Overall, Course 3 (C3) Overall, and All Courses Overall.
Population: Modified intent-to-treat (mITT) population - mITT populations for Courses 1, 2 and 3 were defined as all participants who received the first course, first 2 courses and all 3 courses of treatment respectively. Only participants with a positive ADA status were included in the analysis.
Measure: Number; unit: Percentage of Participants
Groups:
- Rituximab-EU Total: Participants who received Rituximab-EU in the B3281001 study were either assigned Rituximab-EU in the first course of B3281004, or PF-05280586. This measures the total percentage of B3281001 Rituximab-EU participants.
- Rituximab-US Total: Participants who received Rituximab-US in the B3281001 study were either assigned Rituximab-US in the first course of B3281004, or PF-05280586. This measures the total percentage of B3281001 Rituximab-US participants.
Arm/Group | PF-05280586/PF-05280586/PF-05280586 | Rituximab-EU/PF-05280586/PF-05280586 | PF-05280586/PF-05280586/PF-05280586 (EU) | Rituximab-EU Total | Rituximab-US/PF-05280586/PF-05280586 | PF-05280586/PF-05280586/PF-05280586 (US) | Rituximab-US Total
Number analyzed (Participants) | 58 | 32 | 33 | 65 | 30 | 30 | 60
Percentage of Participants
  Total (C1) +ve: number analyzed (Participants) | 57 | 31 | 33 | 64 | 30 | 30 | 60
  Total (C1) +ve | 3.5 | 0.0 | 15.2 | 7.8 | 13.3 | 6.7 | 10.0
  Total (C2) +ve: number analyzed (Participants) | 53 | 30 | 31 | 61 | 29 | 29 | 58
  Total (C2) +ve | 5.7 | 3.3 | 0.0 | 1.6 | 0.0 | 6.9 | 3.4
  Total (C3) +ve: number analyzed (Participants) | 48 | 30 | 30 | 60 | 27 | 29 | 56
  Total (C3) +ve | 2.1 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  C1 to C3 +ve | 8.6 | 3.1 | 15.2 | 9.2 | 13.3 | 6.7 | 10.0

2. Primary Outcome: Percentage of Participants by ADA Status Using Anti-Rituximab Antibody Assay
Description: Serum samples were collected to determine the presence of ADA using two validated assays, one specific for PF-05280586 and one specific for the licensed drug products. For participants assigned to PF-05280586 in Study B3281001, blood samples were screened for ADA using the assay specific to PF-05280586; if the blood samples were confirmed to be positive for ADA against PF-05280586, the samples were also analyzed using the assay specific for the licensed drug products to assess cross-reactivity of the ADA. For participants assigned to the licensed products in Study B3281001, blood samples were screened for ADA using both assays in order to assess any product-specific ADA and/or cross-reactivity for the transition from the licensed products to PF-05280586.
Time Frame: Course 1 Overall, Course 2 Overall, Course 3 Overall, and All Courses Overall.
Population: mITT population - mITT populations for Courses 1, 2 and 3 were defined as all participants who received the first course, first 2 courses and all 3 courses of treatment respectively. Only participants with a positive ADA status were included in the analysis.
Measure: Number; unit: Percentage of Participants
Arm/Group | PF-05280586/PF-05280586/PF-05280586 | Rituximab-EU/PF-05280586/PF-05280586 | PF-05280586/PF-05280586/PF-05280586 (EU) | Rituximab-EU Total | Rituximab-US/PF-05280586/PF-05280586 | PF-05280586/PF-05280586/PF-05280586 (US) | Rituximab-US Total
Number analyzed (Participants) | 58 | 32 | 33 | 65 | 30 | 30 | 60
Percentage of Participants
  Total (C1) +ve: number analyzed (Participants) | 57 | 31 | 33 | 64 | 30 | 30 | 60
  Total (C1) +ve | 3.5 | 3.2 | 15.2 | 9.4 | 10.0 | 10.0 | 10.0
  Total (C2) +ve: number analyzed (Participants) | 53 | 30 | 31 | 61 | 29 | 29 | 58
  Total (C2) +ve | 5.7 | 6.7 | 3.2 | 4.9 | 3.4 | 13.8 | 8.6
  Total (C3) +ve: number analyzed (Participants) | 48 | 30 | 30 | 60 | 27 | 29 | 56
  Total (C3) +ve | 2.1 | 0.0 | 3.3 | 1.7 | 0.0 | 3.4 | 1.8
  C1 to C3 +ve | 8.6 | 6.3 | 18.2 | 12.3 | 13.3 | 13.3 | 13.3

3. Primary Outcome: Percentage of Participants by Neutralizing Antibody (Nab) Status in Participants With a Positive ADA Using Anti-PF-05280586 NAb Assay
Description: Blood samples that were confirmed as positive for ADA were further evaluated for Nab using validated assays - None of the ADA samples tested positive for NAb.
Time Frame: Weeks 1, 3, 13, and 25 (Course 1, Course 2, and Course 3).
Population: mITT Population. Only participants with a positive ADA status were included in the analysis.
Arm/Group | PF-05280586/PF-05280586/PF-05280586 | Rituximab-EU/PF-05280586/PF-05280586 | PF-05280586/PF-05280586/PF-05280586 (EU) | Rituximab-EU Total | Rituximab-US/PF-05280586/PF-05280586 | PF-05280586/PF-05280586/PF-05280586 (US) | Rituximab-US Total
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Percentage of Participants by Nab Status in Participants With a Positive ADA Using Anti-PF-05280586 NAb Assay Using Anti-Rituximab NAb Assay
Description: Blood samples that were confirmed as positive for ADA were further evaluated for Nab using validated assays. - None of the ADA samples tested positive for NAb.
Time Frame: Weeks 1, 3, 13, and 25 (Course 1, Course 2, and Course 3).
Population: mITT Population. Only participants with a positive ADA status were included in the analysis.
Arm/Group | PF-05280586/PF-05280586/PF-05280586 | Rituximab-EU/PF-05280586/PF-05280586 | PF-05280586/PF-05280586/PF-05280586 (EU) | Rituximab-EU Total | Rituximab-US/PF-05280586/PF-05280586 | PF-05280586/PF-05280586/PF-05280586 (US) | Rituximab-US Total
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Mean Rituximab Serum Trough Concentrations
Description: Serum samples for determination of drug concentrations were collected pre-dose concurrent with ADA sample collection. Drug concentrations in the samples were determined using a validated assay.
Time Frame: Weeks 1, 3, 13, and 25 (Course 1, Course 2, and Course 3), Follow up Months 3, 6, 9, and 12. Course 3/Week 25 is End of Treatment (EOT).
Population: mITT Population - mITT populations for Courses 1, 2 and 3 were defined as all participants who received the first course, first 2 courses and all 3 courses of treatment respectively.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter
Arm/Group | PF-05280586/PF-05280586/PF-05280586 | Rituximab-EU/PF-05280586/PF-05280586 | PF-05280586/PF-05280586/PF-05280586 (EU) | Rituximab-US/PF-05280586/PF-05280586 | PF-05280586/PF-05280586/PF-05280586 (US)
Number analyzed (Participants) | 58 | 32 | 33 | 30 | 30
nanograms per milliliter
  Course 1/Week 1: number analyzed (Participants) | 51 | 27 | 31 | 29 | 28
  Course 1/Week 1 | 636.5 (816.33) | 855.5 (1594.51) | 416.6 (615.86) | 1525.8 (3709.90) | 980.0 (2091.41)
  Course 1/Week 3: number analyzed (Participants) | 57 | 31 | 33 | 30 | 30
  Course 1/Week 3 | 103019.3 (29250.13) | 114341.9 (39023.45) | 89790.9 (23247.03) | 96323.3 (33396.81) | 107790.0 (26168.99)
  Course 1/Week 13: number analyzed (Participants) | 56 | 30 | 33 | 30 | 29
  Course 1/Week 13 | 22613.1 (16526.33) | 27542.3 (18879.35) | 16973.6 (10736.22) | 26359.8 (27063.70) | 31006.6 (23055.79)
  Course 1/Week 25: number analyzed (Participants) | 32 | 10 | 20 | 12 | 19
  Course 1/Week 25 | 2844.2 (4271.65) | 3573.3 (3569.90) | 1719.3 (3383.03) | 8205.1 (9923.43) | 3005.6 (5227.33)
  Course 2/Week 1: number analyzed (Participants) | 54 | 30 | 31 | 29 | 29
  Course 2/Week 1 | 1628.2 (2712.30) | 2493.2 (3631.38) | 924.1 (1546.20) | 3463.6 (5311.01) | 3596.1 (5514.43)
  Course 2/Week 3: number analyzed (Participants) | 53 | 30 | 30 | 29 | 27
  Course 2/Week 3 | 108064.2 (37043.94) | 114266.7 (29897.86) | 91006.7 (23725.24) | 102937.9 (29824.58) | 114992.6 (31832.89)
  Course 2/Week 13: number analyzed (Participants) | 52 | 30 | 30 | 29 | 29
  Course 2/Week 13 | 26527.9 (17903.00) | 31829.7 (17954.12) | 21467.0 (11390.72) | 27730.7 (21932.00) | 36007.9 (23651.20)
  Course 2/Week 25: number analyzed (Participants) | 29 | 10 | 18 | 14 | 15
  Course 2/Week 25 | 3431.9 (4155.80) | 4074.2 (5043.55) | 1375.8 (1507.10) | 5103.3 (5344.88) | 5228.6 (7171.47)
  Course 3/Week 1: number analyzed (Participants) | 48 | 30 | 30 | 27 | 29
  Course 3/Week 1 | 3347.7 (6919.26) | 4276.1 (4959.22) | 1569.5 (2592.13) | 3239.2 (4330.47) | 4372.0 (5836.09)
  Course 3/Week 3: number analyzed (Participants) | 48 | 30 | 30 | 27 | 29
  Course 3/Week 3 | 101043.8 (27832.21) | 118256.7 (30549.75) | 96213.3 (22232.76) | 107677.8 (38759.97) | 116134.5 (29028.01)
  Course 3/Week 13: number analyzed (Participants) | 46 | 29 | 29 | 25 | 29
  Course 3/Week 13 | 26795.2 (18635.09) | 31180.0 (20926.62) | 21268.6 (11639.25) | 28801.2 (21593.73) | 33489.7 (21522.53)
  Course 3/Week 25 (EOT): number analyzed (Participants) | 53 | 30 | 31 | 28 | 26
  Course 3/Week 25 (EOT) | 5908.1 (22274.41) | 6485.6 (12462.24) | 6539.7 (23577.35) | 8603.7 (13217.69) | 4887.2 (5543.05)
  Follow up-Month 3: number analyzed (Participants) | 35 | 22 | 21 | 15 | 22
  Follow up-Month 3 | 2448.3 (13132.59) | 9061.5 (30261.67) | 208.3 (255.87) | 2477.5 (5571.32) | 4199.1 (15777.12)
  Follow up-Month 6: number analyzed (Participants) | 29 | 19 | 15 | 9 | 19
  Follow up-Month 6 | 44.2 (140.06) | 99.3 (253.66) | 17.4 (46.39) | 140.8 (297.54) | 4631.8 (19826.17)
  Follow up-Month 9: number analyzed (Participants) | 4 | 0 | 0 | 0 | 2
  Follow up-Month 9 | 0.0 (0.0) |  |  |  | 0.0 (0.0)
  Follow up-Month 12: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1
  Follow up-Month 12 |  |  |  |  | 0.0

6. Primary Outcome: Cluster of Differentiation 19 (CD19+) B Cell Count
Description: Blood samples were assayed for CD19+ B-cell counts using laser scanning cytometry.
Time Frame: Weeks 1, 6, 13, and 25 (Course 1 and Course 2), Weeks 1, 13, 25 (Course 3), and Follow up Months 3, 6, and 9.
Population: as for outcome 5
Measure: Median (Full Range); unit: cells per microliter
Arm/Group | PF-05280586/PF-05280586/PF-05280586 | Rituximab-EU/PF-05280586/PF-05280586 | PF-05280586/PF-05280586/PF-05280586 (EU) | Rituximab-US/PF-05280586/PF-05280586 | PF-05280586/PF-05280586/PF-05280586 (US)
Number analyzed (Participants) | 58 | 32 | 33 | 30 | 30
cells per microliter
  Course 1/Week 1: number analyzed (Participants) | 49 | 28 | 22 | 23 | 25
  Course 1/Week 1 | 0.0 [0.0 to 109.2] | 1.1 [0.0 to 105.6] | 0.6 [0.0 to 55.9] | 0.0 [0.0 to 115.9] | 0.6 [0.0 to 677.5]
  Course 1/Week 6: number analyzed (Participants) | 57 | 28 | 33 | 29 | 28
  Course 1/Week 6 | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 16.7] | 0.0 [0.0 to 0.6] | 0.0 [0.0 to 1.8] | 0.0 [0.0 to 9.2]
  Course 1/Week 13: number analyzed (Participants) | 54 | 31 | 33 | 29 | 27
  Course 1/Week 13 | 0.0 [0.0 to 0.2] | 0.0 [0.0 to 34.9] | 0.0 [0.0 to 4.2] | 0.0 [0.0 to 0.4] | 0.0 [0.0 to 10.3]
  Course 1/Week 25: number analyzed (Participants) | 34 | 10 | 22 | 13 | 18
  Course 1/Week 25 | 0.0 [0.0 to 27.9] | 0.0 [0.0 to 62.7] | 0.0 [0.0 to 67.9] | 0.0 [0.0 to 123.4] | 0.0 [0.0 to 0.0]
  Course 2/Week 1: number analyzed (Participants) | 51 | 29 | 29 | 28 | 28
  Course 2/Week 1 | 0.0 [0.0 to 146.1] | 0.0 [0.0 to 164.0] | 0.0 [0.0 to 77.3] | 0.0 [0.0 to 89.1] | 0.0 [0.0 to 79.8]
  Course 2/Week 6: number analyzed (Participants) | 49 | 30 | 28 | 29 | 27
  Course 2/Week 6 | 0.0 [0.0 to 410.3] | 0.0 [0.0 to 1.5] | 0.0 [0.0 to 13.3] | 0.0 [0.0 to 0.8] | 0.0 [0.0 to 0.5]
  Course 2/Week 13: number analyzed (Participants) | 50 | 28 | 29 | 27 | 29
  Course 2/Week 13 | 0.0 [0.0 to 8.6] | 0.0 [0.0 to 1.7] | 0.0 [0.0 to 13.8] | 0.0 [0.0 to 0.6] | 0.0 [0.0 to 16.7]
  Course 2/Week 25: number analyzed (Participants) | 27 | 9 | 20 | 15 | 15
  Course 2/Week 25 | 0.0 [0.0 to 7.7] | 0.0 [0.0 to 68.4] | 0.0 [0.0 to 11.3] | 0.0 [0.0 to 1.7] | 0.0 [0.0 to 9.6]
  Course 3/Week 1: number analyzed (Participants) | 44 | 29 | 29 | 25 | 27
  Course 3/Week 1 | 0.0 [0.0 to 15.8] | 0.0 [0.0 to 140.1] | 0.0 [0.0 to 25.2] | 0.0 [0.0 to 56.0] | 0.0 [0.0 to 14.3]
  Course 3/Week 13: number analyzed (Participants) | 43 | 28 | 28 | 23 | 24
  Course 3/Week 13 | 0.0 [0.0 to 9.0] | 0.0 [0.0 to 2.4] | 0.0 [0.0 to 1.3] | 0.0 [0.0 to 32.7] | 0.0 [0.0 to 2.7]
  Course 3/Week 25 (EOT): number analyzed (Participants) | 49 | 28 | 30 | 27 | 29
  Course 3/Week 25 (EOT) | 0.0 [0.0 to 23.8] | 0.0 [0.0 to 27.3] | 0.0 [0.0 to 10.1] | 0.0 [0.0 to 321.9] | 0.0 [0.0 to 50.5]
  Follow up-month 3: number analyzed (Participants) | 30 | 19 | 17 | 13 | 19
  Follow up-month 3 | 0.2 [0.0 to 66.5] | 0.0 [0.0 to 60.9] | 1.7 [0.0 to 94.8] | 0.5 [0.0 to 50.2] | 0.0 [0.0 to 211.6]
  Follow up-Month 6: number analyzed (Participants) | 25 | 18 | 14 | 7 | 15
  Follow up-Month 6 | 7.5 [0.0 to 131.6] | 0.4 [0.0 to 124.7] | 6.8 [0.0 to 109.5] | 10.5 [0.0 to 77.3] | 1.1 [0.0 to 177.8]
  Follow up-Month 9: number analyzed (Participants) | 2 | 0 | 0 | 0 | 1
  Follow up-Month 9 | 39.4 [5.0 to 73.9] |  |  |  | 66.3 [66.3 to 66.3]

7. Primary Outcome: Circulating Immunoglobulin G (IgG) Concentrations
Description: Blood samples for immunoglobulin assessments were obtained to determine IgG levels in serum.
Time Frame: Screening, Week 25 (Course 1), and Weeks 1 and 25 (Course 2 and Course 3).
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: grams per liter (g/L)
Arm/Group | PF-05280586/PF-05280586/PF-05280586 | Rituximab-EU/PF-05280586/PF-05280586 | PF-05280586/PF-05280586/PF-05280586 (EU) | Rituximab-US/PF-05280586/PF-05280586 | PF-05280586/PF-05280586/PF-05280586 (US)
Number analyzed (Participants) | 58 | 32 | 33 | 30 | 30
grams per liter (g/L)
  Screening: number analyzed (Participants) | 53 | 30 | 32 | 29 | 30
  Screening | 11.7 (3.06) | 10.9 (2.54) | 11.6 (2.85) | 11.3 (3.12) | 11.8 (3.52)
  Course 1/Week 25: number analyzed (Participants) | 35 | 9 | 22 | 13 | 19
  Course 1/Week 25 | 10.4 (3.20) | 10.7 (3.71) | 11.2 (2.50) | 10.3 (3.50) | 11.4 (3.92)
  Course 2/Week 1: number analyzed (Participants) | 54 | 30 | 31 | 29 | 29
  Course 2/Week 1 | 10.5 (2.73) | 10.2 (2.78) | 10.8 (2.55) | 10.2 (2.29) | 10.9 (3.59)
  Course 2/Week 25: number analyzed (Participants) | 29 | 9 | 20 | 15 | 16
  Course 2/Week 25 | 10.6 (2.85) | 8.9 (2.40) | 10.4 (2.11) | 9.2 (2.00) | 11.4 (4.08)
  Course 3/Week 1: number analyzed (Participants) | 48 | 30 | 30 | 27 | 29
  Course 3/Week 1 | 10.6 (2.92) | 10.2 (2.61) | 10.6 (2.81) | 9.7 (2.44) | 10.3 (3.88)
  Course 3/Week 25 (EOT): number analyzed (Participants) | 54 | 31 | 30 | 29 | 30
  Course 3/Week 25 (EOT) | 10.4 (2.86) | 9.8 (3.04) | 10.3 (2.34) | 9.7 (2.30) | 10.2 (3.25)

8. Primary Outcome: Circulating Immunoglobulin M (IgM) Concentrations
Description: Blood samples for immunoglobulin assessments were obtained to determine IgM levels in serum.
Time Frame: Screening, Week 25 (Course 1), and Weeks 1 and 25 (Course 2 and Course 3).
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | PF-05280586/PF-05280586/PF-05280586 | Rituximab-EU/PF-05280586/PF-05280586 | PF-05280586/PF-05280586/PF-05280586 (EU) | Rituximab-US/PF-05280586/PF-05280586 | PF-05280586/PF-05280586/PF-05280586 (US)
Number analyzed (Participants) | 58 | 32 | 33 | 30 | 30
g/L
  Screening: number analyzed (Participants) | 45 | 22 | 19 | 22 | 23
  Screening | 1.0 (0.50) | 1.1 (0.73) | 1.1 (0.70) | 1.1 (0.79) | 1.0 (0.57)
  Course 1/Week 25: number analyzed (Participants) | 35 | 10 | 22 | 13 | 19
  Course 1/Week 25 | 0.8 (0.47) | 1.1 (0.62) | 0.9 (0.60) | 1.0 (0.72) | 0.9 (0.45)
  Course 2/Week 1: number analyzed (Participants) | 54 | 30 | 31 | 29 | 29
  Course 2/Week 1 | 0.8 (0.48) | 0.9 (0.56) | 0.9 (0.64) | 0.9 (0.61) | 0.8 (0.47)
  Course 2/Week 25: number analyzed (Participants) | 29 | 9 | 20 | 15 | 16
  Course 2/Week 25 | 0.8 (0.55) | 0.8 (0.46) | 0.9 (0.64) | 0.9 (0.63) | 0.8 (0.50)
  Course 3/Week 1: number analyzed (Participants) | 48 | 30 | 30 | 27 | 29
  Course 3/Week 1 | 0.8 (0.43) | 0.8 (0.46) | 0.8 (0.57) | 0.8 (0.52) | 0.7 (0.40)
  Course 3/Week 25 (EOT): number analyzed (Participants) | 54 | 31 | 30 | 29 | 30
  Course 3/Week 25 (EOT) | 0.7 (0.39) | 0.7 (0.44) | 0.8 (0.54) | 0.8 (0.52) | 0.7 (0.38)

9. Primary Outcome: Circulating Rheumatoid Factor (RF) Concentrations
Description: RF is the auto-antibody directed against IgG. Blood samples were obtained to determine RF levels in serum.
Time Frame: Week 1 and 25 (Course 1, Course 2, and Course 3).
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: international units per milliliter
Arm/Group | PF-05280586/PF-05280586/PF-05280586 | Rituximab-EU/PF-05280586/PF-05280586 | PF-05280586/PF-05280586/PF-05280586 (EU) | Rituximab-US/PF-05280586/PF-05280586 | PF-05280586/PF-05280586/PF-05280586 (US)
Number analyzed (Participants) | 58 | 32 | 33 | 30 | 30
international units per milliliter
  Course 1/Week 1: number analyzed (Participants) | 53 | 28 | 31 | 25 | 29
  Course 1/Week 1 | 105.6 (203.88) | 431.3 (1074.13) | 128.7 (201.11) | 75.2 (102.41) | 109.1 (139.79)
  Course 1/Week 25: number analyzed (Participants) | 35 | 10 | 22 | 13 | 19
  Course 1/Week 25 | 56.1 (104.12) | 714.8 (1471.95) | 101.5 (165.85) | 53.2 (59.22) | 66.5 (69.70)
  Course 2/Week 1: number analyzed (Participants) | 54 | 30 | 31 | 29 | 29
  Course 2/Week 1 | 92.6 (181.91) | 279.3 (737.00) | 132.9 (234.84) | 59.5 (76.56) | 58.6 (73.13)
  Course 2/Week 25: number analyzed (Participants) | 29 | 9 | 20 | 15 | 16
  Course 2/Week 25 | 59.5 (117.79) | 448.0 (945.12) | 62.4 (89.14) | 52.0 (54.97) | 44.2 (44.34)
  Course 3/Week 1: number analyzed (Participants) | 48 | 30 | 30 | 27 | 29
  Course 3/Week 1 | 51.7 (89.51) | 217.3 (697.30) | 74.9 (128.83) | 51.8 (92.06) | 40.4 (45.90)
  Course 3/Week 25 (EOT): number analyzed (Participants) | 55 | 31 | 30 | 29 | 30
  Course 3/Week 25 (EOT) | 46.2 (76.85) | 181.2 (551.49) | 57.1 (107.47) | 45.0 (66.43) | 38.2 (41.46)

10. Primary Outcome: Anti-Cyclic Citrullinated Peptide (Anti-CCP) and Complement
Description: Blood samples were obtained to determine anti-CCP and compliment levels in serum.
Time Frame: Week 1 and 25 (Course 1, Course 2, and Course 3).
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: U/mL
Arm/Group | PF-05280586/PF-05280586/PF-05280586 | Rituximab-EU/PF-05280586/PF-05280586 | PF-05280586/PF-05280586/PF-05280586 (EU) | Rituximab-US/PF-05280586/PF-05280586 | PF-05280586/PF-05280586/PF-05280586 (US)
Number analyzed (Participants) | 58 | 32 | 33 | 30 | 30
U/mL
  Course 1/Week 1: number analyzed (Participants) | 54 | 28 | 31 | 26 | 28
  Course 1/Week 1 | 293.7 (206.64) | 346.1 (206.78) | 311.5 (198.13) | 223.9 (224.86) | 306.1 (210.82)
  Course 1/Week 25: number analyzed (Participants) | 34 | 9 | 22 | 11 | 19
  Course 1/Week 25 | 266.9 (222.12) | 230.8 (207.06) | 300.9 (199.02) | 258.0 (227.91) | 263.6 (190.26)
  Course 2/Week 1: number analyzed (Participants) | 54 | 30 | 31 | 29 | 29
  Course 2/Week 1 | 285.7 (211.65) | 305.2 (208.41) | 324.6 (196.92) | 241.5 (229.00) | 262.2 (210.17)
  Course 2/Week 25: number analyzed (Participants) | 29 | 9 | 20 | 15 | 16
  Course 2/Week 25 | 259.0 (224.11) | 332.0 (184.78) | 273.3 (188.63) | 230.1 (232.38) | 237.9 (204.70)
  Course 3/Week 1: number analyzed (Participants) | 48 | 30 | 30 | 27 | 29
  Course 3/Week 1 | 270.0 (213.62) | 290.2 (200.75) | 308.3 (189.51) | 214.3 (228.46) | 234.6 (212.97)
  Course 3/Week 25 (EOT): number analyzed (Participants) | 55 | 30 | 30 | 29 | 30
  Course 3/Week 25 (EOT) | 249.6 (212.37) | 250.4 (190.55) | 265.7 (207.79) | 214.4 (222.43) | 245.1 (207.29)

11. Primary Outcome: Mean Change From Initial Study Baseline in Disease Activity Score (DAS28)-C-Reactive Protein (CRP) - by the End of Course 1
Description: The disease activity score (DAS) assessment is a continuous composite measure derived using differential weighting given to the following 4 components: tender/painful joint count (28 joints), swollen joint count (28 joints), CRP and patient's global assessment of arthritis Visual Analog Scale (VAS). The formula for calculation of DAS28-CRP from these 4 components is DAS28-CRP equals (=) 0.56 square root (sqrt) (DAS 28 tender joint count) + 0.28 sqrt (DAS 28 swollen joint count) + 0.36 natural log [ln] (CRP [milligrams per liter, mg/L] +1) + 0.014 (global assessment of health [GH]) + 0.96. Total score range: 0 to 9.4, higher score indicated more disease activity.
Time Frame: Baseline B3281001, Week 1, 6, 13, and 25 (Course 1).
Population: mITT Population - The mITT population for Course 1 was defined as all participants who received the treatment of the first course of study B3281004.
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- PF-05280586: by the End of Course 1: This treatment group, which received PF-05280586 during the B3281001 study, received IV rituximab (PF-05280586) infusion 1000 mg/500 mL (preceded by 100 mg IV methylprednisolone or its equivalent, an antipyretic, and an antihistamine) on Study Days 1 and 15 of the first 24-week (±8 week) course in this three course study. Participants continued to receive a stable background regimen of methotrexate 10 to 25 mg/week (7.5 mg/week in the event of prior poor tolerance). Folate supplementation was encouraged according to local standard of care.
- Rituximab-EU: by the End of Course 1: This treatment group, which received Rituximab-EU in the B3281001 study, received IV rituximab (MabThera) infusion 1000 mg/500 mL (preceded by 100 mg IV methylprednisolone or its equivalent, an antipyretic, and an antihistamine) on Study Days 1 and 15 of the first 24-week (±8 week) course in this three course study. Participants continued to receive a stable background regimen of methotrexate 10 to 25 mg/week (7.5 mg/week in the event of prior poor tolerance). Folate supplementation was encouraged according to local standard of care.
- PF-05280586 (EU): by the End of Course 1: This treatment group, which received Rituximab-EU in the B3281001 study, received IV rituximab (PF-05280586) infusion 1000 mg/500 mL (preceded by 100 mg IV methylprednisolone or its equivalent, an antipyretic, and an antihistamine) on Study Days 1 and 15 of the first 24-week (±8 week) course in this three course study. Participants continued to receive a stable background regimen of methotrexate 10 to 25 mg/week (7.5 mg/week in the event of prior poor tolerance). Folate supplementation was encouraged according to local standard of care.
- Rituximab-US: by the End of Course 1: This treatment group, which received Rituximab-US in the B3281001 study, received IV rituximab (Rituxan) infusion 1000 mg/500 mL (preceded by 100 mg methylprednisolone or its equivalent, an antipyretic, and an antihistamine) on Study Days 1 and 15 of the first 24-week (±8 week) course in this three course study. Participants continued to receive a stable background regimen of methotrexate 10 to 25 mg/week (7.5 mg/week in the event of prior poor tolerance) for up to 25 weeks. Folate supplementation was encouraged according to local standard of care.
- PF-05280586 (US): by the End of Course 1: This treatment group, which received Rituximab-US in the B3281001 study, received IV rituximab (PF-05280586) infusion 1000 mg/500 mL (preceded by 100 mg IV methylprednisolone or its equivalent, an antipyretic, and an antihistamine) on Study Days 1 and 15 of the first 24-week (±8 week) course in this three course study. Participants continued to receive a stable background regimen of methotrexate 10 to 25 mg/week (7.5 mg/week in the event of prior poor tolerance). Folate supplementation was encouraged according to local standard of care.
Arm/Group | PF-05280586: by the End of Course 1 | Rituximab-EU: by the End of Course 1 | PF-05280586 (EU): by the End of Course 1 | Rituximab-US: by the End of Course 1 | PF-05280586 (US): by the End of Course 1
Number analyzed (Participants) | 58 | 32 | 33 | 30 | 30
Units on a scale
  Baseline B3281001 | 5.59 (0.862) | 5.81 (0.926) | 5.80 (0.988) | 6.16 (0.870) | 6.12 (0.784)
  Change at Course 1/Week 1: number analyzed (Participants) | 51 | 28 | 31 | 25 | 28
  Change at Course 1/Week 1 | -1.24 (1.126) | -1.86 (1.223) | -1.94 (1.315) | -2.02 (1.508) | -1.95 (1.211)
  Change at Course 1/Week 6: number analyzed (Participants) | 56 | 31 | 32 | 30 | 28
  Change at Course 1/Week 6 | -2.03 (1.378) | -2.59 (1.088) | -2.54 (1.322) | -2.50 (1.454) | -2.66 (1.226)
  Change at Course 1/Week 13: number analyzed (Participants) | 56 | 30 | 33 | 29 | 29
  Change at Course 1/Week 13 | -2.37 (1.134) | -2.78 (1.355) | -2.66 (1.439) | -2.85 (1.368) | -2.76 (1.200)
  Change at Course 1/Week 25: number analyzed (Participants) | 35 | 10 | 22 | 13 | 19
  Change at Course 1/Week 25 | -2.35 (1.310) | -2.32 (1.166) | -2.24 (1.182) | -2.15 (1.109) | -2.50 (1.179)

12. Primary Outcome: Mean Change From Initial Study Baseline in Disease Activity Score (DAS28)-C-Reactive Protein (CRP) - by the End of Course 2
Description: as for outcome 11
Time Frame: Baseline B3281001, Week 1, 6, 13, and 25 (Course 1 and Course 2).
Population: mITT Population - The mITT population for Course 2 was defined as all participants who received the treatments of the first 2 courses of study B3281004.
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- PF-05280586: by the End of Course 2: This treatment group, which received PF-05280586 in the B3281001 study, received IV rituximab (PF-05280586) infusion 1000 mg/500 mL (preceded by 100 mg IV methylprednisolone or its equivalent, an antipyretic, and an antihistamine) on Study Days 1 and 15 of the first two 24-week (±8 week) courses in this three course study. Participants continued to receive a stable background regimen of methotrexate 10 to 25 mg/week (7.5 mg/week in the event of prior poor tolerance). Folate supplementation was encouraged according to local standard of care.
- Rituximab-EU/PF-05280586: by the End of Course 2: This treatment group, which received Rituximab-EU in the B3281001 study, received IV rituximab (MabThera) infusion 1000 mg/500 mL (preceded by 100 mg IV methylprednisolone or its equivalent, an antipyretic, and an antihistamine) on Study Days 1 and 15 of the first 24-week (±8 week) course in this three course study, followed by IV rituximab (PF-05280586) infusion 1000 mg/500 mL (preceded by 100 mg IV methylprednisolone or its equivalent, an antipyretic, and an antihistamine) on Study Days 1 and 15 of the second 24-week (±8 week) course. Participants continued to receive a stable background regimen of methotrexate 10 to 25 mg/week (7.5 mg/week in the event of prior poor tolerance). Folate supplementation was encouraged according to local standard of care.
- PF-05280586 (EU): by the End of Course 2: This treatment group, which received Rituximab-EU in the B3281001 study, received IV rituximab (PF-05280586) infusion 1000 mg/500 mL (preceded by 100 mg IV methylprednisolone or its equivalent, an antipyretic, and an antihistamine) on Study Days 1 and 15 of the first two 24-week (±8 week) courses in this three course study. Participants continued to receive a stable background regimen of methotrexate 10 to 25 mg/week (7.5 mg/week in the event of prior poor tolerance). Folate supplementation was encouraged according to local standard of care.
- Rituximab-US/PF-05280586: by the End of Course 2: This treatment group, which received Rituximab-US in the B3281001 study, received IV rituximab (Rituxan) infusion 1000 mg/500 mL (preceded by 100 mg methylprednisolone or its equivalent, an antipyretic, and an antihistamine) on Study Days 1 and 15 of the first 24-week (±8 week) course in this three course study, followed by IV rituximab (PF-05280586) infusion 1000 mg/500 mL (preceded by 100 mg IV methylprednisolone or its equivalent, an antipyretic, and an antihistamine) on Study Days 1 and 15 of the second 24-week (±8 week) course. Participants continued to receive a stable background regimen of methotrexate 10 to 25 mg/week (7.5 mg/week in the event of prior poor tolerance) for up to 25 weeks. Folate supplementation was encouraged according to local standard of care.
- PF-05280586 (US): by the End of Course 2: This treatment group, which received Rituximab-US in the B3281001 study, received IV rituximab (PF-05280586) infusion 1000 mg/500 mL (preceded by 100 mg IV methylprednisolone or its equivalent, an antipyretic, and an antihistamine) on Study Days 1 and 15 of the first two 24-week (±8 week) courses in this three course study. Participants continued to receive a stable background regimen of methotrexate 10 to 25 mg/week (7.5 mg/week in the event of prior poor tolerance). Folate supplementation was encouraged according to local standard of care.
Arm/Group | PF-05280586: by the End of Course 2 | Rituximab-EU/PF-05280586: by the End of Course 2 | PF-05280586 (EU): by the End of Course 2 | Rituximab-US/PF-05280586: by the End of Course 2 | PF-05280586 (US): by the End of Course 2
Number analyzed (Participants) | 54 | 30 | 31 | 29 | 29
Units on a scale
  Baseline B3281001 | 5.59 (0.893) | 5.81 (0.956) | 5.77 (1.009) | 6.13 (0.865) | 6.10 (0.792)
  Change at Course 1/Week 1: number analyzed (Participants) | 49 | 26 | 29 | 24 | 27
  Change at Course 1/Week 1 | -1.27 (1.120) | -1.82 (1.257) | -1.92 (1.147) | -1.93 (1.466) | -1.99 (1.218)
  Change at Course 1/Week 6: number analyzed (Participants) | 53 | 30 | 30 | 29 | 27
  Change at Course 1/Week 6 | -2.11 (1.353) | -2.56 (1.091) | -2.53 (1.205) | -2.44 (1.441) | -2.71 (1.211)
  Change at Course 1/Week 13: number analyzed (Participants) | 54 | 30 | 31 | 28 | 29
  Change at Course 1/Week 13 | -2.41 (1.110) | -2.78 (1.355) | -2.67 (1.315) | -2.76 (1.318) | -2.76 (1.200)
  Change at Course 1/Week 25: number analyzed (Participants) | 35 | 10 | 20 | 12 | 19
  Change at Course 1/Week 25 | -2.35 (1.310) | -2.32 (1.166) | -2.19 (1.034) | -2.02 (1.038) | -2.50 (1.179)
  Change at Course 2/Week 1 | -1.98 (1.480) | -2.05 (1.275) | -1.92 (1.132) | -2.20 (1.295) | -2.34 (1.036)
  Change at Course 2/Week 6: number analyzed (Participants) | 52 | 29 | 29 | 29 | 29
  Change at Course 2/Week 6 | -2.66 (1.177) | -2.74 (1.552) | -2.75 (1.148) | -2.92 (1.231) | -3.00 (1.089)
  Change at Course 2/Week 13: number analyzed (Participants) | 52 | 29 | 30 | 27 | 29
  Change at Course 2/Week 13 | -2.35 (1.319) | -2.56 (1.644) | -2.65 (1.113) | -2.88 (1.476) | -3.21 (1.135)
  Change at Course 2/Week 25: number analyzed (Participants) | 29 | 9 | 20 | 15 | 16
  Change at Course 2/Week 25 | -2.30 (1.061) | -3.14 (1.013) | -2.42 (1.125) | -2.35 (1.010) | -2.82 (0.901)

13. Primary Outcome: Mean Change From Initial Study Baseline in Disease Activity Score (DAS28)-C-Reactive Protein (CRP) - by the End of Course 3
Description: as for outcome 11
Time Frame: Baseline B3281001, Week 1, 6, 13, and 25 (Course 1 and Course 2), and Week 1, 13, and 25 (Course 3).
Population: mITT Population - The mITT population for Course 3 was defined as all participants who received the treatments of all 3 courses of study B3281004.
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- PF-05280586: by the End of Course 3: This treatment group, which received PF-05280586 in the B3281001 study, received IV rituximab (PF-05280586) infusion 1000 mg/500 mL (preceded by 100 mg IV methylprednisolone or its equivalent, an antipyretic, and an antihistamine) on Study Days 1 and 15 of all three 24-week (±8 week) courses in this three course study. Participants continued to receive a stable background regimen of methotrexate 10 to 25 mg/week (7.5 mg/week in the event of prior poor tolerance). Folate supplementation was encouraged according to local standard of care.
- Rituximab-EU/PF-05280586/PF-05280586: by the End of Course 3: This treatment group, which received Rituximab-EU in the B3281001 study, received IV rituximab (MabThera) infusion 1000 mg/500 mL (preceded by 100 mg IV methylprednisolone or its equivalent, an antipyretic, and an antihistamine) on Study Days 1 and 15 of the first 24-week (±8 week) course in this three course study, followed by IV rituximab (PF-05280586) infusion 1000 mg/500 mL (preceded by 100 mg IV methylprednisolone or its equivalent, an antipyretic, and an antihistamine) on Study Days 1 and 15 of the second and third 24-week (±8 week) courses. Participants continued to receive a stable background regimen of methotrexate 10 to 25 mg/week (7.5 mg/week in the event of prior poor tolerance). Folate supplementation was encouraged according to local standard of care.
- PF-05280586 (EU): by the End of Course 3: This treatment group, which received Rituximab-EU in the B3281001 study, received IV rituximab (PF-05280586) infusion 1000 mg/500 mL (preceded by 100 mg IV methylprednisolone or its equivalent, an antipyretic, and an antihistamine) on Study Days 1 and 15 of all three 24-week (±8 week) courses in this three course study. Participants continued to receive a stable background regimen of methotrexate 10 to 25 mg/week (7.5 mg/week in the event of prior poor tolerance). Folate supplementation was encouraged according to local standard of care.
- Rituximab-US/PF-05280586/PF-05280586: by the End of Course 3: This treatment group, which received Rituximab-US in the B3281001 study, received IV rituximab (Rituxan) infusion 1000 mg/500 mL (preceded by 100 mg methylprednisolone or its equivalent, an antipyretic, and an antihistamine) on Study Days 1 and 15 of the first 24-week (±8 week) course in this three course study, followed by IV rituximab (PF-05280586) infusion 1000 mg/500 mL (preceded by 100 mg IV methylprednisolone or its equivalent, an antipyretic, and an antihistamine) on Study Days 1 and 15 of the second and third 24-week (±8 week) courses. Participants continued to receive a stable background regimen of methotrexate 10 to 25 mg/week (7.5 mg/week in the event of prior poor tolerance) for up to 25 weeks. Folate supplementation was encouraged according to local standard of care.
- PF-05280586 (US): by the End of Course 3: This treatment group, which received Rituximab-US in the B3281001 study, received IV rituximab (PF-05280586) infusion 1000 mg/500 mL (preceded by 100 mg IV methylprednisolone or its equivalent, an antipyretic, and an antihistamine) on Study Days 1 and 15 of all three 24-week (±8 week) courses in this three course study. Participants continued to receive a stable background regimen of methotrexate 10 to 25 mg/week (7.5 mg/week in the event of prior poor tolerance). Folate supplementation was encouraged according to local standard of care.
Arm/Group | PF-05280586: by the End of Course 3 | Rituximab-EU/PF-05280586/PF-05280586: by the End of Course 3 | PF-05280586 (EU): by the End of Course 3 | Rituximab-US/PF-05280586/PF-05280586: by the End of Course 3 | PF-05280586 (US): by the End of Course 3
Number analyzed (Participants) | 48 | 30 | 30 | 27 | 29
Units on a scale
  Baseline B3281001 | 5.54 (0.896) | 5.81 (0.956) | 5.79 (1.019) | 6.14 (0.886) | 6.10 (0.792)
  Change at Course 1/Week 1: number analyzed (Participants) | 44 | 26 | 28 | 23 | 27
  Change at Course 1/Week 1 | -1.25 (1.158) | -1.82 (1.257) | -1.86 (1.121) | -2.01 (1.438) | -1.99 (1.218)
  Change at Course 1/Week 6: number analyzed (Participants) | 47 | 30 | 29 | 27 | 27
  Change at Course 1/Week 6 | -2.10 (1.380) | -2.56 (1.091) | -2.51 (1.221) | -2.53 (1.438) | -2.71 (1.211)
  Change at Course 1/Week 13: number analyzed (Participants) | 48 | 30 | 30 | 26 | 29
  Change at Course 1/Week 13 | -2.47 (1.101) | -2.78 (1.355) | -2.64 (1.322) | -2.82 (1.284) | -2.76 (1.200)
  Change at Course 1/Week 25: number analyzed (Participants) | 32 | 10 | 19 | 11 | 19
  Change at Course 1/Week 25 | -2.25 (1.293) | -2.32 (1.166) | -2.12 (1.023) | -2.21 (0.848) | -2.50 (1.179)
  Change at Course 2/Week 1 | -1.93 (1.500) | -2.05 (1.275) | -1.87 (1.118) | -2.27 (1.314) | -2.34 (1.036)
  Change at Course 2/Week 6: number analyzed (Participants) | 47 | 29 | 29 | 27 | 29
  Change at Course 2/Week 6 | -2.62 (1.172) | -2.74 (1.552) | -2.75 (1.148) | -2.97 (1.241) | -3.00 (1.089)
  Change at Course 2/Week 13: number analyzed (Participants) | 47 | 29 | 30 | 25 | 29
  Change at Course 2/Week 13 | -2.34 (1.369) | -2.56 (1.644) | -2.65 (1.113) | -2.96 (1.507) | -3.21 (1.135)
  Change at Course 2/Week 25: number analyzed (Participants) | 26 | 9 | 20 | 14 | 16
  Change at Course 2/Week 25 | -2.34 (1.114) | -3.14 (1.013) | -2.42 (1.125) | -2.41 (1.020) | -2.82 (0.901)
  Change at Course 3/Week 1 | -1.98 (1.477) | -2.34 (1.525) | -2.33 (1.106) | -2.43 (1.600) | -2.51 (1.238)
  Change at Course 3/Week 13: number analyzed (Participants) | 46 | 30 | 29 | 25 | 29
  Change at Course 3/Week 13 | -2.46 (1.428) | -2.78 (1.519) | -2.74 (1.103) | -3.09 (1.489) | -3.03 (1.145)
  Change at Course 3/Week 25: number analyzed (Participants) | 47 | 29 | 29 | 27 | 29
  Change at Course 3/Week 25 | -2.30 (1.245) | -2.53 (1.641) | -2.59 (1.314) | -2.88 (1.127) | -2.86 (1.392)

14. Primary Outcome: Percentage of Participants With Good European League Against Rheumatism (EULAR) Response Based on DAS28 - by the End of Course 1
Description: The DAS28-based EULAR response criteria were used to measure individual response as none, good, and moderate, depending on the extent of change from baseline and the level of disease activity reached. Good responders had a change from baseline greater than (>) 1.2 with present DAS28 less than or equal to (≤) 3.2; moderate responders had a change from baseline >0.6 and ≤1.2 with present DAS28 ≤3.2 or change from baseline >0.6 with present DAS28 >3.2 and ≤5.1 or change from baseline >1.2 with present DAS28 >5.1; non-responders had a change from baseline ≤0.6 with present DAS28 ≤5.1 or change from baseline ≤1.2 with present DAS28 >5.1.
Time Frame: Week 1, 6, 13, and 25 (Course 1).
Population: as for outcome 11
Measure: Number; unit: Percentage of Participants
Arm/Group | PF-05280586: by the End of Course 1 | Rituximab-EU: by the End of Course 1 | PF-05280586 (EU): by the End of Course 1 | Rituximab-US: by the End of Course 1 | PF-05280586 (US): by the End of Course 1
Number analyzed (Participants) | 58 | 32 | 33 | 30 | 30
Percentage of Participants
  Course 1/Week 1: number analyzed (Participants) | 51 | 28 | 31 | 25 | 28
  Course 1/Week 1 | 13.7 | 25.0 | 32.3 | 32.0 | 21.4
  Course 1/Week 6: number analyzed (Participants) | 56 | 31 | 32 | 30 | 28
  Course 1/Week 6 | 35.7 | 54.8 | 46.9 | 43.3 | 46.4
  Course 1/Week 13: number analyzed (Participants) | 56 | 30 | 33 | 29 | 29
  Course 1/Week 13 | 51.8 | 66.7 | 51.5 | 44.8 | 44.8
  Course 1/Week 25: number analyzed (Participants) | 35 | 10 | 22 | 13 | 19
  Course 1/Week 25 | 57.1 | 20.0 | 36.4 | 23.1 | 36.8

15. Primary Outcome: Percentage of Participants With Good European League Against Rheumatism (EULAR) Response Based on DAS28 - by the End of Course 2
Description: as for outcome 14
Time Frame: Week 1, 6, 13, and 25 (Course 1 and Course 2).
Population: as for outcome 12
Measure: Number; unit: Percentage of Participants
Arm/Group | PF-05280586: by the End of Course 2 | Rituximab-EU/PF-05280586: by the End of Course 2 | PF-05280586 (EU): by the End of Course 2 | Rituximab-US/PF-05280586: by the End of Course 2 | PF-05280586 (US): by the End of Course 2
Number analyzed (Participants) | 54 | 30 | 31 | 29 | 29
Percentage of Participants
  Course 1/Week 1: number analyzed (Participants) | 49 | 26 | 29 | 24 | 27
  Course 1/Week 1 | 14.3 | 26.9 | 31.0 | 29.2 | 22.2
  Course 1/Week 6: number analyzed (Participants) | 53 | 30 | 30 | 29 | 27
  Course 1/Week 6 | 37.7 | 53.3 | 46.7 | 41.4 | 48.1
  Course 1/Week 13: number analyzed (Participants) | 54 | 30 | 31 | 28 | 29
  Course 1/Week 13 | 51.9 | 66.7 | 51.6 | 42.9 | 44.8
  Course 1/Week 25: number analyzed (Participants) | 35 | 10 | 20 | 12 | 19
  Course 1/Week 25 | 57.1 | 20.0 | 35.0 | 25.0 | 36.8
  Course 2/Week 1 | 44.4 | 33.3 | 29.0 | 27.6 | 24.1
  Course 2/Week 6: number analyzed (Participants) | 52 | 29 | 29 | 29 | 29
  Course 2/Week 6 | 61.5 | 55.2 | 51.7 | 37.9 | 48.3
  Course 2/Week 13: number analyzed (Participants) | 52 | 29 | 30 | 27 | 29
  Course 2/Week 13 | 51.9 | 51.7 | 53.3 | 55.6 | 65.5
  Course 2/Week 25: number analyzed (Participants) | 29 | 9 | 20 | 15 | 16
  Course 2/Week 25 | 55.2 | 66.7 | 50.0 | 46.7 | 43.8

16. Primary Outcome: Percentage of Participants With Good European League Against Rheumatism (EULAR) Response Based on DAS28 - by the End of Course 3
Description: as for outcome 14
Time Frame: Week 1, 6, 13, and 25 (Course 1 and Course 2) and Week 1, 13, and 25 (Course 3).
Population: as for outcome 13
Measure: Number; unit: Percentage of Participants
Arm/Group | PF-05280586: by the End of Course 3 | Rituximab-EU/PF-05280586/PF-05280586: by the End of Course 3 | PF-05280586 (EU): by the End of Course 3 | Rituximab-US/PF-05280586/PF-05280586: by the End of Course 3 | PF-05280586 (US): by the End of Course 3
Number analyzed (Participants) | 48 | 30 | 30 | 27 | 29
Percentage of Participants
  Course 1/Week 1: number analyzed (Participants) | 44 | 26 | 28 | 23 | 27
  Course 1/Week 1 | 15.9 | 26.9 | 28.6 | 30.4 | 22.2
  Course 1/Week 6: number analyzed (Participants) | 47 | 30 | 29 | 27 | 27
  Course 1/Week 6 | 40.4 | 53.3 | 44.8 | 44.4 | 48.1
  Course 1/Week 13: number analyzed (Participants) | 48 | 30 | 30 | 26 | 29
  Course 1/Week 13 | 56.3 | 66.7 | 50.0 | 42.3 | 44.8
  Course 1/Week 25: number analyzed (Participants) | 32 | 10 | 19 | 11 | 19
  Course 1/Week 25 | 53.1 | 20.0 | 31.6 | 27.3 | 36.8
  Course 2/Week 1 | 47.9 | 33.3 | 26.7 | 29.6 | 24.1
  Course 2/Week 6: number analyzed (Participants) | 47 | 29 | 29 | 27 | 29
  Course 2/Week 6 | 59.6 | 55.2 | 51.7 | 40.7 | 48.3
  Course 2/Week 13: number analyzed (Participants) | 47 | 29 | 30 | 25 | 29
  Course 2/Week 13 | 51.1 | 51.7 | 53.3 | 60.0 | 65.5
  Course 2/Week 25: number analyzed (Participants) | 26 | 9 | 20 | 14 | 16
  Course 2/Week 25 | 57.7 | 66.7 | 50.0 | 50.0 | 43.8
  Course 3/Week 1 | 43.8 | 43.3 | 36.7 | 37.0 | 34.5
  Course 3/Week 13: number analyzed (Participants) | 46 | 30 | 29 | 25 | 29
  Course 3/Week 13 | 56.5 | 53.3 | 58.6 | 60.0 | 58.6
  Course 3/Week 25 (EOT): number analyzed (Participants) | 47 | 29 | 29 | 27 | 29
  Course 3/Week 25 (EOT) | 48.9 | 48.3 | 55.2 | 48.1 | 51.7

17. Primary Outcome: Percentage of Participants With Low Disease Activity State (LDAS) (≤3.2) - by the End of Course 1
Description: The DAS assessment is a continuous composite measure derived using differential weighting given to the following 4 components: tender/painful joint count (28 joints), swollen joint count (28 joints), CRP and patient's global assessment of arthritis VAS. The formula for calculation of DAS28-CRP from these 4 components is DAS28-CRP = 0.56 sqrt (DAS 28 tender joint count) + 0.28 sqrt (DAS 28 swollen joint count) + 0.36 (ln CRP [mg/L] +1) + 0.014 (GH) + 0.96. Total score range: 0 to 9.4, higher score indicated more disease activity. DAS28-CRP ≤3.2 implied low disease activity.
Time Frame: Week 1, 6, 13, and 25 (Course 1).
Population: as for outcome 11
Measure: Number; unit: Percentage of Participants
Arm/Group | PF-05280586: by the End of Course 1 | Rituximab-EU: by the End of Course 1 | PF-05280586 (EU): by the End of Course 1 | Rituximab-US: by the End of Course 1 | PF-05280586 (US): by the End of Course 1
Number analyzed (Participants) | 58 | 32 | 33 | 30 | 30
Percentage of Participants
  Course 1/Week 1: number analyzed (Participants) | 51 | 28 | 31 | 25 | 28
  Course 1/Week 1 | 13.7 | 25.0 | 32.3 | 32.0 | 21.4
  Course 1/Week 6: number analyzed (Participants) | 56 | 31 | 32 | 30 | 28
  Course 1/Week 6 | 35.7 | 54.8 | 50.0 | 43.3 | 46.4
  Course 1/Week 13: number analyzed (Participants) | 56 | 30 | 33 | 29 | 29
  Course 1/Week 13 | 51.8 | 66.7 | 57.6 | 44.8 | 44.8
  Course 1/Week 25: number analyzed (Participants) | 35 | 10 | 22 | 13 | 19
  Course 1/Week 25 | 57.1 | 20.0 | 45.5 | 23.1 | 36.8

18. Primary Outcome: Percentage of Participants With Low Disease Activity State (LDAS) (≤3.2) - by the End of Course 2
Description: as for outcome 17
Time Frame: Week 1, 6, 13, and 25 (Course 1 and Course 2).
Population: as for outcome 12
Measure: Number; unit: Percentage of Participants
Arm/Group | PF-05280586: by the End of Course 2 | Rituximab-EU/PF-05280586: by the End of Course 2 | PF-05280586 (EU): by the End of Course 2 | Rituximab-US/PF-05280586: by the End of Course 2 | PF-05280586 (US): by the End of Course 2
Number analyzed (Participants) | 54 | 30 | 31 | 29 | 29
Percentage of Participants
  Course 1/Week 1: number analyzed (Participants) | 49 | 26 | 29 | 24 | 27
  Course 1/Week 1 | 14.3 | 26.9 | 31.0 | 29.2 | 22.2
  Course 1/Week 6: number analyzed (Participants) | 53 | 30 | 30 | 29 | 27
  Course 1/Week 6 | 37.7 | 53.3 | 50.0 | 41.4 | 48.1
  Course 1/Week 13: number analyzed (Participants) | 54 | 30 | 31 | 28 | 29
  Course 1/Week 13 | 51.9 | 66.7 | 58.1 | 42.9 | 44.8
  Course 1/Week 25: number analyzed (Participants) | 35 | 10 | 20 | 12 | 19
  Course 1/Week 25 | 57.1 | 20.0 | 45.0 | 25.0 | 36.8
  Course 2/Week 1 | 44.4 | 33.3 | 29.0 | 27.6 | 24.1
  Course 2/Week 6: number analyzed (Participants) | 52 | 29 | 29 | 29 | 29
  Course 2/Week 6 | 61.5 | 55.2 | 55.2 | 37.9 | 48.3
  Course 2/Week 13: number analyzed (Participants) | 52 | 29 | 30 | 27 | 29
  Course 2/Week 13 | 51.9 | 51.7 | 56.7 | 55.6 | 65.5
  Course 2/Week 25: number analyzed (Participants) | 29 | 9 | 20 | 15 | 16
  Course 2/Week 25 | 55.2 | 66.7 | 50.0 | 46.7 | 43.8

19. Primary Outcome: Percentage of Participants With Low Disease Activity State (LDAS) (≤3.2) - by the End of Course 3
Description: as for outcome 17
Time Frame: Week 1, 6, 13, and 25 (Course 1 and Course 2), and Week 1, 13, and 25 (Course 3).
Population: as for outcome 13
Measure: Number; unit: Percentage of Participants
Arm/Group | PF-05280586: by the End of Course 3 | Rituximab-EU/PF-05280586/PF-05280586: by the End of Course 3 | PF-05280586 (EU): by the End of Course 3 | Rituximab-US/PF-05280586/PF-05280586: by the End of Course 3 | PF-05280586 (US): by the End of Course 3
Number analyzed (Participants) | 48 | 30 | 30 | 27 | 29
Percentage of Participants
  Course 1/Week 1: number analyzed (Participants) | 44 | 26 | 28 | 23 | 27
  Course 1/Week 1 | 15.9 | 26.9 | 28.6 | 30.4 | 22.2
  Course 1/Week 6: number analyzed (Participants) | 47 | 30 | 29 | 27 | 27
  Course 1/Week 6 | 40.4 | 53.3 | 48.3 | 44.4 | 48.1
  Course 1/Week 13: number analyzed (Participants) | 48 | 30 | 30 | 26 | 29
  Course 1/Week 13 | 56.3 | 66.7 | 56.7 | 42.3 | 44.8
  Course 1/Week 25: number analyzed (Participants) | 32 | 10 | 19 | 11 | 19
  Course 1/Week 25 | 53.1 | 20.0 | 42.1 | 27.3 | 36.8
  Course 2/Week 1 | 47.9 | 33.3 | 26.7 | 29.6 | 24.1
  Course 2/Week 6: number analyzed (Participants) | 47 | 29 | 29 | 27 | 29
  Course 2/Week 6 | 59.6 | 55.2 | 55.2 | 40.7 | 48.3
  Course 2/Week 13: number analyzed (Participants) | 47 | 29 | 30 | 25 | 29
  Course 2/Week 13 | 51.1 | 51.7 | 56.7 | 60.0 | 65.5
  Course 2/Week 25: number analyzed (Participants) | 26 | 9 | 20 | 14 | 16
  Course 2/Week 25 | 57.7 | 66.7 | 50.0 | 50.0 | 43.8
  Course 3/Week 1 | 43.8 | 43.3 | 40.0 | 37.0 | 34.5
  Course 3/Week 13: number analyzed (Participants) | 46 | 30 | 29 | 25 | 29
  Course 3/Week 13 | 58.7 | 56.7 | 58.6 | 60.0 | 58.6
  Course 3/Week 25 (EOT): number analyzed (Participants) | 47 | 29 | 29 | 27 | 29
  Course 3/Week 25 (EOT) | 48.9 | 48.3 | 58.6 | 48.1 | 51.7

20. Primary Outcome: Percentage of Participants With DAS Remission (DAS28-CRP Less Than [<] 2.6) - by the End of Course 1
Description: The DAS assessment is a continuous composite measure derived using differential weighting given to the following 4 components: tender/painful joint count (28 joints), swollen joint count (28 joints), CRP and patient's global assessment of arthritis VAS. The formula for calculation of DAS28-CRP from these 4 components is DAS28-CRP = 0.56 sqrt (DAS 28 tender joint count) + 0.28 sqrt (DAS 28 swollen joint count) + 0.36 (ln CRP [mg/L] +1) + 0.014 (GH) + 0.96. Total score range: 0 to 9.4, higher score indicated more disease activity. DAS28-CRP <2.6 implied remission.
Time Frame: Week 1, 6, 13, and 25 (Course 1).
Population: as for outcome 11
Measure: Number; unit: Percentage of Participants
Arm/Group | PF-05280586: by the End of Course 1 | Rituximab-EU: by the End of Course 1 | PF-05280586 (EU): by the End of Course 1 | Rituximab-US: by the End of Course 1 | PF-05280586 (US): by the End of Course 1
Number analyzed (Participants) | 58 | 32 | 33 | 30 | 30
Percentage of Participants
  Course 1/Week 1: number analyzed (Participants) | 51 | 28 | 31 | 25 | 28
  Course 1/Week 1 | 3.9 | 10.7 | 19.4 | 12.0 | 7.1
  Course 1/Week 6: number analyzed (Participants) | 56 | 31 | 32 | 30 | 28
  Course 1/Week 6 | 32.1 | 38.7 | 34.4 | 30.0 | 32.1
  Course 1/Week 13: number analyzed (Participants) | 56 | 30 | 33 | 29 | 29
  Course 1/Week 13 | 33.9 | 46.7 | 45.5 | 27.6 | 37.9
  Course 1/Week 25: number analyzed (Participants) | 35 | 10 | 22 | 13 | 19
  Course 1/Week 25 | 45.7 | 20.0 | 27.3 | 15.4 | 21.1

21. Primary Outcome: Percentage of Participants With DAS Remission (DAS28-CRP Less Than [<] 2.6) - by the End of Course 2
Description: as for outcome 20
Time Frame: Week 1, 6, 13, and 25 (Course 1 and Course 2).
Population: as for outcome 12
Measure: Number; unit: Percentage of Participants
Arm/Group | PF-05280586: by the End of Course 2 | Rituximab-EU/PF-05280586: by the End of Course 2 | PF-05280586 (EU): by the End of Course 2 | Rituximab-US/PF-05280586: by the End of Course 2 | PF-05280586 (US): by the End of Course 2
Number analyzed (Participants) | 54 | 30 | 31 | 29 | 29
Percentage of Participants
  Course 1/Week 1: number analyzed (Participants) | 49 | 26 | 29 | 24 | 27
  Course 1/Week 1 | 4.1 | 11.5 | 17.2 | 12.5 | 7.4
  Course 1/Week 6: number analyzed (Participants) | 53 | 30 | 30 | 29 | 27
  Course 1/Week 6 | 34.0 | 36.7 | 33.3 | 31.0 | 33.3
  Course 1/Week 13: number analyzed (Participants) | 54 | 30 | 31 | 28 | 29
  Course 1/Week 13 | 35.2 | 46.7 | 45.2 | 25.0 | 37.9
  Course 1/Week 25: number analyzed (Participants) | 35 | 10 | 20 | 12 | 19
  Course 1/Week 25 | 45.7 | 20.0 | 25.0 | 16.7 | 21.1
  Course 2/Week 1 | 22.2 | 13.3 | 19.4 | 17.2 | 10.3
  Course 2/Week 6: number analyzed (Participants) | 52 | 29 | 29 | 29 | 29
  Course 2/Week 6 | 42.3 | 41.4 | 24.1 | 37.9 | 31.0
  Course 2/Week 13: number analyzed (Participants) | 52 | 29 | 30 | 27 | 29
  Course 2/Week 13 | 30.8 | 37.9 | 33.3 | 33.3 | 44.8
  Course 2/Week 25: number analyzed (Participants) | 29 | 9 | 20 | 15 | 16
  Course 2/Week 25 | 27.6 | 33.3 | 35.0 | 20.0 | 25.0

22. Primary Outcome: Percentage of Participants With DAS Remission (DAS28-CRP Less Than [<] 2.6) - by the End of Course 3
Description: as for outcome 20
Time Frame: Week 1, 6, 13, and 25 (Course 1 and Course 2), and Week 1, 13, and 25 (Course 3).
Population: as for outcome 13
Measure: Number; unit: Percentage of Participants
Arm/Group | PF-05280586: by the End of Course 3 | Rituximab-EU/PF-05280586/PF-05280586: by the End of Course 3 | PF-05280586 (EU): by the End of Course 3 | Rituximab-US/PF-05280586/PF-05280586: by the End of Course 3 | PF-05280586 (US): by the End of Course 3
Number analyzed (Participants) | 48 | 30 | 30 | 27 | 29
Percentage of Participants
  Course 1/Week 1: number analyzed (Participants) | 44 | 26 | 28 | 23 | 27
  Course 1/Week 1 | 4.5 | 11.5 | 14.3 | 13.0 | 7.4
  Course 1/Week 6: number analyzed (Participants) | 47 | 30 | 29 | 27 | 27
  Course 1/Week 6 | 36.2 | 36.7 | 31.0 | 33.3 | 33.3
  Course 1/Week 13: number analyzed (Participants) | 48 | 30 | 30 | 26 | 29
  Course 1/Week 13 | 39.6 | 46.7 | 43.3 | 26.9 | 37.9
  Course 1/Week 25: number analyzed (Participants) | 32 | 10 | 19 | 11 | 19
  Course 1/Week 25 | 43.8 | 20.0 | 21.1 | 18.2 | 21.1
  Course 2/Week 1 | 22.9 | 13.3 | 16.7 | 18.5 | 10.3
  Course 2/Week 6: number analyzed (Participants) | 47 | 29 | 29 | 27 | 29
  Course 2/Week 6 | 44.7 | 41.4 | 24.1 | 40.7 | 31.0
  Course 2/Week 13: number analyzed (Participants) | 47 | 29 | 30 | 25 | 29
  Course 2/Week 13 | 29.8 | 37.9 | 33.3 | 36.0 | 44.8
  Course 2/Week 25: number analyzed (Participants) | 26 | 9 | 20 | 14 | 16
  Course 2/Week 25 | 30.8 | 33.3 | 35.0 | 21.4 | 25.0
  Course 3/Week 1 | 22.9 | 30.0 | 26.7 | 22.2 | 24.1
  Course 3/Week 13: number analyzed (Participants) | 46 | 30 | 29 | 25 | 29
  Course 3/Week 13 | 41.3 | 46.7 | 44.8 | 44.0 | 34.5
  Course 3/Week 25 (EOT): number analyzed (Participants) | 47 | 29 | 29 | 27 | 29
  Course 3/Week 25 (EOT) | 34.0 | 37.9 | 41.4 | 33.3 | 37.9

23. Primary Outcome: Percentage of Participants With American College of Rheumatology (ACR) 20% Improvement (ACR20) Response - by the End of Course 1
Description: ACR20 response: ≥ 20 percent (%) improvement in tender/painful joint count; ≥ 20% improvement in swollen joint count; and ≥ 20% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of arthritis pain; participant global assessment of arthritis; physician global assessment of arthritis; self-assessed disability (disability index of the Health Assessment Questionnaire [HAQ]); and CRP.
Time Frame: Week 1, 6, 13, and 25 (Course 1).
Population: as for outcome 11
Measure: Number; unit: Percentage of participants
Arm/Group | PF-05280586: by the End of Course 1 | Rituximab-EU: by the End of Course 1 | PF-05280586 (EU): by the End of Course 1 | Rituximab-US: by the End of Course 1 | PF-05280586 (US): by the End of Course 1
Number analyzed (Participants) | 58 | 32 | 33 | 30 | 30
Percentage of participants
  Course 1/Week 1 | 50.0 | 59.4 | 63.6 | 66.7 | 60.0
  Course 1/Week 6: number analyzed (Participants) | 57 | 31 | 33 | 30 | 30
  Course 1/Week 6 | 66.7 | 71.0 | 84.8 | 73.3 | 76.7
  Course 1/Week 13: number analyzed (Participants) | 56 | 31 | 33 | 30 | 29
  Course 1/Week 13 | 69.6 | 77.4 | 84.8 | 83.3 | 82.8
  Course 1/Week 25: number analyzed (Participants) | 35 | 10 | 22 | 13 | 19
  Course 1/Week 25 | 77.1 | 90.0 | 81.8 | 76.9 | 73.7

24. Primary Outcome: Percentage of Participants With American College of Rheumatology (ACR) 20% Improvement (ACR20) Response - by the End of Course 2
Description: as for outcome 23
Time Frame: Week 1, 6, 13, and 25 (Course 1 and Course 2).
Population: as for outcome 12
Measure: Number; unit: Percentage of participants
Arm/Group | PF-05280586: by the End of Course 2 | Rituximab-EU/PF-05280586: by the End of Course 2 | PF-05280586 (EU): by the End of Course 2 | Rituximab-US/PF-05280586: by the End of Course 2 | PF-05280586 (US): by the End of Course 2
Number analyzed (Participants) | 54 | 30 | 31 | 29 | 29
Percentage of participants
  Course 1/Week 1 | 51.9 | 60.0 | 64.5 | 65.5 | 62.1
  Course 1/Week 6 | 70.4 | 70.0 | 87.1 | 72.4 | 75.9
  Course 1/Week 13 | 70.4 | 76.7 | 87.1 | 82.8 | 82.8
  Course 1/Week 25: number analyzed (Participants) | 35 | 10 | 20 | 12 | 19
  Course 1/Week 25 | 77.1 | 90.0 | 80.0 | 75.0 | 73.7
  Course 2/Week 1 | 66.7 | 63.3 | 71.0 | 72.4 | 69.0
  Course 2/Week 6: number analyzed (Participants) | 53 | 30 | 29 | 29 | 29
  Course 2/Week 6 | 79.2 | 70.0 | 93.1 | 79.3 | 86.2
  Course 2/Week 13: number analyzed (Participants) | 53 | 30 | 30 | 28 | 29
  Course 2/Week 13 | 66.0 | 60.0 | 86.7 | 78.6 | 89.7
  Course 2/Week 25: number analyzed (Participants) | 29 | 9 | 20 | 15 | 16
  Course 2/Week 25 | 79.3 | 88.9 | 85.0 | 80.0 | 93.8

25. Primary Outcome: Percentage of Participants With American College of Rheumatology (ACR) 20% Improvement (ACR20) Response - by the End of Course 3
Description: as for outcome 23
Time Frame: Week 1, 6, 13, and 25 (Course 1 and Course 2), and Week 1, 13, and 25 (Course 3).
Population: as for outcome 13
Measure: Number; unit: Percentage of participants
Arm/Group | PF-05280586: by the End of Course 3 | Rituximab-EU/PF-05280586/PF-05280586: by the End of Course 3 | PF-05280586 (EU): by the End of Course 3 | Rituximab-US/PF-05280586/PF-05280586: by the End of Course 3 | PF-05280586 (US): by the End of Course 3
Number analyzed (Participants) | 48 | 30 | 30 | 27 | 29
Percentage of participants
  Course 1/Week 1 | 50.0 | 60.0 | 63.3 | 70.4 | 62.1
  Course 1/Week 6 | 70.8 | 70.0 | 86.7 | 74.1 | 75.9
  Course 1/Week 13 | 70.8 | 76.7 | 86.7 | 85.2 | 82.8
  Course 1/Week 25: number analyzed (Participants) | 32 | 10 | 19 | 11 | 19
  Course 1/Week 25 | 75.0 | 90.0 | 78.9 | 81.8 | 73.7
  Course 2/Week 1 | 68.8 | 63.3 | 70.0 | 74.1 | 69.0
  Course 2/Week 6: number analyzed (Participants) | 48 | 30 | 29 | 27 | 29
  Course 2/Week 6 | 77.1 | 70.0 | 93.1 | 81.5 | 86.2
  Course 2/Week 13: number analyzed (Participants) | 48 | 30 | 30 | 26 | 29
  Course 2/Week 13 | 64.6 | 60.0 | 86.7 | 76.9 | 89.7
  Course 2/Week 25: number analyzed (Participants) | 26 | 9 | 20 | 14 | 16
  Course 2/Week 25 | 80.8 | 88.9 | 85.0 | 85.7 | 93.8
  Course 3/Week 1 | 60.4 | 56.7 | 70.0 | 59.3 | 69.0
  Course 3/Week 13: number analyzed (Participants) | 46 | 30 | 29 | 26 | 29
  Course 3/Week 13 | 67.4 | 73.3 | 82.8 | 69.2 | 82.8
  Course 3/Week 25 (EOT): number analyzed (Participants) | 47 | 30 | 29 | 27 | 29
  Course 3/Week 25 (EOT) | 59.6 | 66.7 | 89.7 | 74.1 | 86.2

26. Primary Outcome: Percentage of Participants With American College of Rheumatology (ACR) 50% Improvement (ACR50) Response - by the End of Course 1
Description: ACR50 response: ≥50% improvement in tender/painful joint count; ≥50% improvement in swollen joint count; and ≥50% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of arthritis pain; participant global assessment of arthritis; physician global assessment of arthritis; self-assessed disability (disability index of the HAQ); and CRP.
Time Frame: Week 1, 6, 13, and 25 (Course 1).
Population: as for outcome 11
Measure: Number; unit: Percentage of Participants
Arm/Group | PF-05280586: by the End of Course 1 | Rituximab-EU: by the End of Course 1 | PF-05280586 (EU): by the End of Course 1 | Rituximab-US: by the End of Course 1 | PF-05280586 (US): by the End of Course 1
Number analyzed (Participants) | 58 | 32 | 33 | 30 | 30
Percentage of Participants
  Course 1/Week 1 | 17.2 | 28.1 | 48.5 | 30.0 | 30.0
  Course 1/Week 6: number analyzed (Participants) | 57 | 31 | 33 | 30 | 30
  Course 1/Week 6 | 33.3 | 51.6 | 51.5 | 50.0 | 53.3
  Course 1/Week 13: number analyzed (Participants) | 56 | 31 | 33 | 30 | 29
  Course 1/Week 13 | 37.5 | 41.9 | 66.7 | 66.7 | 58.6
  Course 1/Week 25: number analyzed (Participants) | 35 | 10 | 22 | 13 | 19
  Course 1/Week 25 | 51.4 | 30.0 | 63.6 | 46.2 | 36.8

27. Primary Outcome: Percentage of Participants With American College of Rheumatology (ACR) 50% Improvement (ACR50) Response - by the End of Course 2
Description: as for outcome 26
Time Frame: Week 1, 6, 13, and 25 (Course 1 and Course 2).
Population: as for outcome 12
Measure: Number; unit: Percentage of Participants
Arm/Group | PF-05280586: by the End of Course 2 | Rituximab-EU/PF-05280586: by the End of Course 2 | PF-05280586 (EU): by the End of Course 2 | Rituximab-US/PF-05280586: by the End of Course 2 | PF-05280586 (US): by the End of Course 2
Number analyzed (Participants) | 54 | 30 | 31 | 29 | 29
Percentage of Participants
  Course 1/Week 1 | 18.5 | 26.7 | 48.4 | 27.6 | 31.0
  Course 1/Week 6 | 35.2 | 50.0 | 51.6 | 48.3 | 55.2
  Course 1/Week 13 | 38.9 | 40.0 | 67.7 | 65.5 | 58.6
  Course 1/Week 25: number analyzed (Participants) | 35 | 10 | 20 | 12 | 19
  Course 1/Week 25 | 51.4 | 30.0 | 65.0 | 41.7 | 36.8
  Course 2/Week 1 | 40.7 | 33.3 | 41.9 | 34.5 | 24.1
  Course 2/Week 6: number analyzed (Participants) | 53 | 30 | 29 | 29 | 29
  Course 2/Week 6 | 50.9 | 53.3 | 58.6 | 55.2 | 55.2
  Course 2/Week 13: number analyzed (Participants) | 53 | 30 | 30 | 28 | 29
  Course 2/Week 13 | 47.2 | 46.7 | 56.7 | 53.6 | 55.2
  Course 2/Week 25: number analyzed (Participants) | 29 | 9 | 20 | 15 | 16
  Course 2/Week 25 | 58.6 | 55.6 | 50.0 | 40.0 | 50.0

28. Primary Outcome: Percentage of Participants With American College of Rheumatology (ACR) 50% Improvement (ACR50) Response - by the End of Course 3
Description: as for outcome 26
Time Frame: Week 1, 6, 13, and 25 (Course 1 and Course 2), and Week 1, 13, and 25 (Course 3).
Population: as for outcome 13
Measure: Number; unit: Percentage of Participants
Arm/Group | PF-05280586: by the End of Course 3 | Rituximab-EU/PF-05280586/PF-05280586: by the End of Course 3 | PF-05280586 (EU): by the End of Course 3 | Rituximab-US/PF-05280586/PF-05280586: by the End of Course 3 | PF-05280586 (US): by the End of Course 3
Number analyzed (Participants) | 48 | 30 | 30 | 27 | 29
Percentage of Participants
  Course 1/Week 1 | 18.8 | 26.7 | 46.7 | 29.6 | 31.0
  Course 1/Week 6 | 33.3 | 50.0 | 50.0 | 51.9 | 55.2
  Course 1/Week 13 | 43.8 | 40.0 | 66.7 | 66.7 | 58.6
  Course 1/Week 25: number analyzed (Participants) | 32 | 10 | 19 | 11 | 19
  Course 1/Week 25 | 46.9 | 30.0 | 63.2 | 45.5 | 36.8
  Course 2/Week 1 | 41.7 | 33.3 | 40.0 | 37.0 | 24.1
  Course 2/Week 6: number analyzed (Participants) | 48 | 30 | 29 | 27 | 29
  Course 2/Week 6 | 50.0 | 53.3 | 58.6 | 55.6 | 55.2
  Course 2/Week 13: number analyzed (Participants) | 48 | 30 | 30 | 26 | 29
  Course 2/Week 13 | 45.8 | 46.7 | 56.7 | 57.7 | 55.2
  Course 2/Week 25: number analyzed (Participants) | 26 | 9 | 20 | 14 | 16
  Course 2/Week 25 | 65.4 | 55.6 | 50.0 | 42.9 | 50.0
  Course 3/Week 1 | 31.3 | 43.3 | 33.3 | 44.4 | 37.9
  Course 3/Week 13: number analyzed (Participants) | 46 | 30 | 29 | 26 | 29
  Course 3/Week 13 | 58.7 | 56.7 | 58.6 | 53.8 | 62.1
  Course 3/Week 25 (EOT): number analyzed (Participants) | 47 | 30 | 29 | 27 | 29
  Course 3/Week 25 (EOT) | 42.6 | 43.3 | 62.1 | 59.3 | 62.1

29. Primary Outcome: Percentage of Participants With American College of Rheumatology (ACR) 70% Improvement (ACR70) Response - by the End of Course 1
Description: ACR70 response: ≥70% improvement in tender/painful joint count; ≥70% improvement in swollen joint count; and ≥70% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of arthritis pain; participant global assessment of arthritis; physician global assessment of arthritis; self-assessed disability (disability index of the HAQ); and CRP.
Time Frame: Week 1, 6, 13, and 25 (Course 1).
Population: as for outcome 11
Measure: Number; unit: Percentage of Participants
Arm/Group | PF-05280586: by the End of Course 1 | Rituximab-EU: by the End of Course 1 | PF-05280586 (EU): by the End of Course 1 | Rituximab-US: by the End of Course 1 | PF-05280586 (US): by the End of Course 1
Number analyzed (Participants) | 58 | 32 | 33 | 30 | 30
Percentage of Participants
  Course 1/Week 1 | 5.2 | 12.5 | 21.2 | 16.7 | 10.0
  Course 1/Week 6: number analyzed (Participants) | 57 | 31 | 33 | 30 | 30
  Course 1/Week 6 | 21.1 | 22.6 | 33.3 | 26.7 | 30.0
  Course 1/Week 13: number analyzed (Participants) | 56 | 31 | 33 | 30 | 29
  Course 1/Week 13 | 23.2 | 32.3 | 36.4 | 33.3 | 34.5
  Course 1/Week 25: number analyzed (Participants) | 35 | 10 | 22 | 13 | 19
  Course 1/Week 25 | 22.9 | 10.0 | 36.4 | 0.0 | 15.8

30. Primary Outcome: Percentage of Participants With American College of Rheumatology (ACR) 70% Improvement (ACR70) Response - by the End of Course 2
Description: as for outcome 29
Time Frame: Week 1, 6, 13, and 25 (Course 1 and Course 2).
Population: as for outcome 12
Measure: Number; unit: Percentage of Participants
Arm/Group | PF-05280586: by the End of Course 2 | Rituximab-EU/PF-05280586: by the End of Course 2 | PF-05280586 (EU): by the End of Course 2 | Rituximab-US/PF-05280586: by the End of Course 2 | PF-05280586 (US): by the End of Course 2
Number analyzed (Participants) | 54 | 30 | 31 | 29 | 29
Percentage of Participants
  Course 1/Week 1 | 5.6 | 10.0 | 19.4 | 13.8 | 10.3
  Course 1/Week 6 | 22.2 | 20.0 | 32.3 | 24.1 | 31.0
  Course 1/Week 13 | 24.1 | 30.0 | 35.5 | 31.0 | 34.5
  Course 1/Week 25: number analyzed (Participants) | 35 | 10 | 20 | 12 | 19
  Course 1/Week 25 | 22.9 | 10.0 | 35.0 | 0.0 | 15.8
  Course 2/Week 1 | 13.0 | 16.7 | 19.4 | 17.2 | 10.3
  Course 2/Week 6: number analyzed (Participants) | 53 | 30 | 29 | 29 | 29
  Course 2/Week 6 | 26.4 | 30.0 | 37.9 | 24.1 | 24.1
  Course 2/Week 13: number analyzed (Participants) | 53 | 30 | 30 | 28 | 29
  Course 2/Week 13 | 30.2 | 30.0 | 33.3 | 32.1 | 24.1
  Course 2/Week 25: number analyzed (Participants) | 29 | 9 | 20 | 15 | 16
  Course 2/Week 25 | 24.1 | 22.2 | 30.0 | 20.0 | 31.3

31. Primary Outcome: Percentage of Participants With American College of Rheumatology (ACR) 70% Improvement (ACR70) Response - by the End of Course 3
Description: as for outcome 29
Time Frame: Week 1, 6, 13, and 25 (Course 1 and Course 2), and Week 1, 13, and 25 (Course 3).
Population: as for outcome 13
Measure: Number; unit: Percentage of Participants
Arm/Group | PF-05280586: by the End of Course 3 | Rituximab-EU/PF-05280586/PF-05280586: by the End of Course 3 | PF-05280586 (EU): by the End of Course 3 | Rituximab-US/PF-05280586/PF-05280586: by the End of Course 3 | PF-05280586 (US): by the End of Course 3
Number analyzed (Participants) | 48 | 30 | 30 | 27 | 29
Percentage of Participants
  Course 1/Week 1 | 6.3 | 10.0 | 16.7 | 14.8 | 10.3
  Course 1/Week 6 | 22.9 | 20.0 | 30.0 | 25.9 | 31.0
  Course 1/Week 13 | 27.1 | 30.0 | 33.3 | 33.3 | 34.5
  Course 1/Week 25: number analyzed (Participants) | 32 | 10 | 19 | 11 | 19
  Course 1/Week 25 | 21.9 | 10.0 | 31.6 | 0.0 | 15.8
  Course 2/Week 1 | 12.5 | 16.7 | 16.7 | 18.5 | 10.3
  Course 2/Week 6: number analyzed (Participants) | 48 | 30 | 29 | 27 | 29
  Course 2/Week 6 | 27.1 | 30.0 | 37.9 | 25.9 | 24.1
  Course 2/Week 13: number analyzed (Participants) | 48 | 30 | 30 | 26 | 29
  Course 2/Week 13 | 29.2 | 30.0 | 33.3 | 34.6 | 24.1
  Course 2/Week 25: number analyzed (Participants) | 26 | 9 | 20 | 14 | 16
  Course 2/Week 25 | 26.9 | 22.2 | 30.0 | 21.4 | 31.3
  Course 3/Week 1 | 12.5 | 23.3 | 20.0 | 33.3 | 20.7
  Course 3/Week 13: number analyzed (Participants) | 48 | 30 | 29 | 26 | 29
  Course 3/Week 13 | 30.4 | 33.3 | 37.9 | 42.3 | 34.5
  Course 3/Week 25 (EOT): number analyzed (Participants) | 47 | 30 | 29 | 27 | 29
  Course 3/Week 25 (EOT) | 25.5 | 20.0 | 34.5 | 37.0 | 24.1

32. Primary Outcome: Percent Change From Initial Study Baseline in Individual Components of the ACR Response: Tender/Painful Joint Count - by the End of Course 1
Description: Sixty-eight joints were assessed by a blinded joint assessor to determine the number of joints that were considered tender or painful. For consistency, a single assessor was preferred to perform all evaluations across the study for an individual participant. The response to pressure/motion on each joint was assessed using the following scale: Present/Absent/Not Done/Not Applicable (to be used for artificial or missing joints). Artificial joints were not be assessed.
Time Frame: Screening, Week 1, 6, 13, and 25 (Course 1).
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Percent change in joint count
Arm/Group | PF-05280586: by the End of Course 1 | Rituximab-EU: by the End of Course 1 | PF-05280586 (EU): by the End of Course 1 | Rituximab-US: by the End of Course 1 | PF-05280586 (US): by the End of Course 1
Number analyzed (Participants) | 58 | 32 | 33 | 30 | 30
Percent change in joint count
  Change at Screening: number analyzed (Participants) | 58 | 32 | 32 | 30 | 30
  Change at Screening | -52.2 (31.46) | -57.1 (37.14) | -64.2 (29.79) | -57.0 (39.55) | -55.2 (31.97)
  Change at Course 1/Week 1 | -41.4 (46.10) | -51.1 (44.62) | -57.8 (40.25) | -50.5 (44.08) | -51.6 (33.00)
  Change at Course 1/Week 6: number analyzed (Participants) | 57 | 31 | 33 | 30 | 30
  Change at Course 1/Week 6 | -52.2 (117.76) | -72.1 (29.69) | -72.5 (31.75) | -68.7 (36.39) | -69.5 (37.71)
  Change at Course 1/Week 13: number analyzed (Participants) | 56 | 31 | 33 | 30 | 29
  Change at Course 1/Week 13 | -70.2 (41.21) | -76.6 (32.37) | -72.9 (28.99) | -70.6 (37.69) | -68.7 (33.16)
  Change at Course 1/Week 25: number analyzed (Participants) | 35 | 10 | 22 | 13 | 19
  Change at Course 1/Week 25 | -52.2 (31.46) | -57.1 (37.14) | -64.2 (29.79) | -57.0 (39.55) | -55.2 (31.97)

33. Primary Outcome: Percent Change From Initial Study Baseline in Individual Components of the ACR Response: Tender/Painful Joint Count - by the End of Course 2
Description: as for outcome 32
Time Frame: Screening, Week 1, 6, 13, and 25 (Course 1 and Course 2).
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Percent change in joint count
Arm/Group | PF-05280586: by the End of Course 2 | Rituximab-EU/PF-05280586: by the End of Course 2 | PF-05280586 (EU): by the End of Course 2 | Rituximab-US/PF-05280586: by the End of Course 2 | PF-05280586 (US): by the End of Course 2
Number analyzed (Participants) | 54 | 30 | 31 | 29 | 29
Percent change in joint count
  Change at Screening: number analyzed (Participants) | 54 | 30 | 30 | 29 | 29
  Change at Screening | -54.1 (31.00) | -56.0 (38.11) | -64.7 (28.61) | -55.5 (39.39) | -55.9 (32.29)
  Change at Course 1/Week 1 | -42.7 (46.01) | -48.9 (45.19) | -57.8 (40.07) | -49.1 (44.15) | -51.9 (33.54)
  Change at Course 1/Week 6 | -53.4 (120.45) | -71.5 (29.97) | -74.1 (29.12) | -67.8 (36.66) | -70.5 (37.95)
  Change at Course 1/Week 13 | -70.9 (40.98) | -75.8 (32.62) | -74.5 (25.85) | -69.6 (37.93) | -68.7 (33.16)
  Change at Course 1/Week 25: number analyzed (Participants) | 35 | 10 | 20 | 12 | 19
  Change at Course 1/Week 25 | -70.7 (34.48) | -74.0 (19.08) | -70.3 (26.87) | -49.8 (44.90) | -69.9 (20.36)
  Change at Course 2/Week 1 | -54.6 (68.22) | -61.5 (30.90) | -60.0 (39.43) | -55.4 (38.38) | -60.0 (30.18)
  Change at Course 2/Week 6: number analyzed (Participants) | 53 | 30 | 29 | 29 | 29
  Change at Course 2/Week 6 | -81.5 (24.73) | -73.7 (31.95) | -79.5 (25.12) | -70.1 (32.79) | -77.3 (27.37)
  Change at Course 2/Week 13: number analyzed (Participants) | 53 | 30 | 30 | 28 | 29
  Change at Course 2/Week 13 | -70.7 (35.12) | -69.3 (39.85) | -77.5 (22.83) | -74.4 (34.04) | -82.5 (21.63)
  Change at Course 2/Week 25: number analyzed (Participants) | 29 | 9 | 20 | 15 | 16
  Change at Course 2/Week 25 | -76.5 (19.30) | -84.9 (19.60) | -72.4 (25.01) | -69.7 (27.10) | -75.5 (14.06)

34. Primary Outcome: Percent Change From Initial Study Baseline in Individual Components of the ACR Response: Tender/Painful Joint Count - by the End of Course 3
Description: as for outcome 32
Time Frame: Screening, Week 1, 6, 13, and 25 (Course 1 and Course 2), and Screening, Week 1, 13, and 25 (Course 3).
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Percent change in joint count
Arm/Group | PF-05280586: by the End of Course 3 | Rituximab-EU/PF-05280586/PF-05280586: by the End of Course 3 | PF-05280586 (EU): by the End of Course 3 | Rituximab-US/PF-05280586/PF-05280586: by the End of Course 3 | PF-05280586 (US): by the End of Course 3
Number analyzed (Participants) | 48 | 30 | 30 | 27 | 29
Percent change in joint count
  Change at Screening: number analyzed (Participants) | 48 | 30 | 29 | 27 | 29
  Change at Screening | -53.4 (31.93) | -56.0 (38.11) | -63.5 (28.31) | -59.6 (37.63) | -55.9 (32.29)
  Change at Course 1/Week 1 | -41.5 (47.81) | -48.9 (45.19) | -56.4 (39.97) | -53.7 (41.95) | -51.9 (33.54)
  Change at Course 1/Week 6 | -53.6 (127.05) | -71.5 (29.97) | -73.3 (29.22) | -72.4 (33.42) | -70.5 (37.95)
  Change at Course 1/Week 13 | -75.1 (30.47) | -75.8 (32.62) | -73.7 (25.85) | -74.4 (28.15) | -68.7 (33.16)
  Change at Course 1/Week 25: number analyzed (Participants) | 32 | 10 | 19 | 11 | 19
  Change at Course 1/Week 25 | -69.0 (35.57) | -74.0 (19.08) | -68.8 (26.66) | -58.9 (33.62) | -69.9 (20.36)
  Change at Course 2/Week 1 | -54.9 (69.76) | -61.5 (30.90) | -58.7 (39.38) | -59.2 (36.67) | -60.0 (30.18)
  Change at Course 2/Week 6: number analyzed (Participants) | 48 | 30 | 29 | 27 | 29
  Change at Course 2/Week 6 | -81.5 (25.65) | -73.7 (31.95) | -79.5 (25.12) | -73.2 (30.50) | -77.3 (27.37)
  Change at Course 2/Week 13: number analyzed (Participants) | 48 | 30 | 30 | 26 | 29
  Change at Course 2/Week 13 | -69.4 (36.44) | -69.3 (39.85) | -77.5 (22.83) | -76.0 (34.73) | -82.5 (21.63)
  Change at Course 2/Week 25: number analyzed (Participants) | 26 | 9 | 20 | 14 | 16
  Change at Course 2/Week 25 | -75.7 (19.82) | -84.9 (19.60) | -72.4 (25.01) | -72.8 (25.18) | -75.5 (14.06)
  Change at Course 3/Week 1 | -57.3 (63.73) | -65.6 (32.53) | -66.5 (30.69) | -59.5 (41.25) | -67.8 (26.58)
  Change at Course 3/Week 13: number analyzed (Participants) | 46 | 30 | 29 | 26 | 29
  Change at Course 3/Week 13 | -69.1 (54.91) | -69.2 (52.97) | -79.6 (22.21) | -80.8 (21.63) | -79.6 (22.11)
  Change at Course 3/Week 25: number analyzed (Participants) | 47 | 30 | 29 | 27 | 29
  Change at Course 3/Week 25 | -71.8 (31.20) | -59.2 (80.64) | -75.6 (29.79) | -79.0 (17.65) | -78.6 (24.11)

35. Primary Outcome: Percent Change From Initial Study Baseline in Individual Components of the ACR Response: Swollen Joint Count - by the End of Course 1
Description: Sixty-six joints were assessed by a blinded joint assessor for swelling. For consistency, a single assessor was preferred to perform all evaluations across the study for an individual participant. The response was assessed using the following scale: Present/Absent/Not Done/Not Applicable (to be used for artificial or missing joints). Artificial joints were not be assessed.
Time Frame: Screening, Week 1, 6, 13, and 25 (Course 1).
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Percent change in joint count
Arm/Group | PF-05280586: by the End of Course 1 | Rituximab-EU: by the End of Course 1 | PF-05280586 (EU): by the End of Course 1 | Rituximab-US: by the End of Course 1 | PF-05280586 (US): by the End of Course 1
Number analyzed (Participants) | 58 | 32 | 33 | 30 | 30
Percent change in joint count
  Change at Screening: number analyzed (Participants) | 58 | 32 | 32 | 30 | 30
  Change at Screening | -58.1 (33.22) | -54.2 (39.43) | -62.9 (32.45) | -54.9 (41.05) | -59.1 (29.43)
  Change at Course 1/Week 1 | -51.7 (40.21) | -49.9 (46.14) | -53.4 (48.36) | -47.9 (55.08) | -58.4 (32.65)
  Change at Course 1/Week 6: number analyzed (Participants) | 57 | 31 | 33 | 30 | 30
  Change at Course 1/Week 6 | -60.2 (116.58) | -55.1 (94.22) | -70.6 (35.20) | -68.2 (45.65) | -76.9 (26.79)
  Change at Course 1/Week 13: number analyzed (Participants) | 56 | 31 | 33 | 30 | 29
  Change at Course 1/Week 13 | -78.0 (29.20) | -47.2 (133.31) | -75.6 (34.36) | -79.5 (22.58) | -70.0 (44.41)
  Change at Course 1/Week 25: number analyzed (Participants) | 35 | 10 | 22 | 13 | 19
  Change at Course 1/Week 25 | -75.0 (27.92) | -74.1 (16.33) | -74.7 (27.15) | -58.6 (50.63) | -67.2 (28.49)

36. Primary Outcome: Percent Change From Initial Study Baseline in Individual Components of the ACR Response: Swollen Joint Count - by the End of Course 2
Description: as for outcome 35
Time Frame: Screening, Week 1, 6, 13, and 25 (Course 1 and Course 2).
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Percent change in joint count
Arm/Group | PF-05280586: by the End of Course 2 | Rituximab-EU/PF-05280586: by the End of Course 2 | PF-05280586 (EU): by the End of Course 2 | Rituximab-US/PF-05280586: by the End of Course 2 | PF-05280586 (US): by the End of Course 2
Number analyzed (Participants) | 54 | 30 | 31 | 29 | 29
Percent change in joint count
  Change at Screening: number analyzed (Participants) | 54 | 30 | 30 | 29 | 29
  Change at Screening | -60.4 (29.31) | -52.5 (40.15) | -64.0 (30.26) | -53.3 (40.86) | -60.2 (29.30)
  Change at Course 1/Week 1 | -55.1 (35.01) | -47.7 (46.81) | -53.8 (48.02) | -46.4 (55.43) | -59.2 (32.91)
  Change at Course 1/Week 6 | -62.7 (117.28) | -53.8 (95.58) | -72.5 (32.18) | -67.2 (46.15) | -78.2 (26.25)
  Change at Course 1/Week 13 | -78.3 (29.13) | -45.4 (135.23) | -77.8 (30.83) | -78.7 (22.64) | -70.0 (44.41)
  Change at Course 1/Week 25: number analyzed (Participants) | 35 | 10 | 20 | 12 | 19
  Change at Course 1/Week 25 | -75.0 (27.92) | -74.1 (16.33) | -76.0 (25.18) | -55.9 (51.86) | -67.2 (28.49)
  Change at Course 2/Week 1 | -58.0 (76.91) | -51.0 (54.16) | -53.1 (46.17) | -59.2 (39.14) | -56.2 (45.29)
  Change at Course 2/Week 6: number analyzed (Participants) | 53 | 30 | 29 | 29 | 29
  Change at Course 2/Week 6 | -81.3 (25.98) | -64.6 (51.49) | -82.3 (21.43) | -74.3 (32.10) | -82.0 (20.56)
  Change at Course 2/Week 13: number analyzed (Participants) | 53 | 30 | 30 | 28 | 29
  Change at Course 2/Week 13 | -77.3 (30.10) | -54.7 (91.62) | -75.0 (34.02) | -76.7 (29.58) | -81.3 (26.43)
  Change at Course 2/Week 25: number analyzed (Participants) | 29 | 9 | 20 | 15 | 16
  Change at Course 2/Week 25 | -75.0 (26.74) | -84.4 (16.09) | -77.9 (21.66) | -77.1 (28.22) | -80.0 (21.86)

37. Primary Outcome: Percent Change From Initial Study Baseline in Individual Components of the ACR Response: Swollen Joint Count - by the End of Course 3
Description: as for outcome 35
Time Frame: Screening, Week 1, 6, 13, and 25 (Course 1 and Course 2), and Screening, Week 1, 13, and 25 (Course 3).
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Percent change in joint count
Arm/Group | PF-05280586: by the End of Course 3 | Rituximab-EU/PF-05280586/PF-05280586: by the End of Course 3 | PF-05280586 (EU): by the End of Course 3 | Rituximab-US/PF-05280586/PF-05280586: by the End of Course 3 | PF-05280586 (US): by the End of Course 3
Number analyzed (Participants) | 48 | 30 | 30 | 27 | 29
Percent change in joint count
  Change at Screening: number analyzed (Participants) | 48 | 30 | 29 | 27 | 29
  Change at Screening | -60.5 (30.41) | -52.5 (40.15) | -62.7 (30.01) | -53.9 (42.34) | -60.2 (29.30)
  Change at Course 1/Week 1 | -55.6 (36.38) | -47.7 (46.81) | -52.2 (48.06) | -49.0 (55.86) | -59.2 (32.91)
  Change at Course 1/Week 6 | -62.1 (124.10) | -53.8 (95.58) | -71.5 (32.31) | -68.2 (47.40) | -78.2 (26.25)
  Change at Course 1/Week 13 | -79.3 (27.17) | -45.4 (135.23) | -77.0 (31.08) | -79.2 (22.12) | -70.0 (44.41)
  Change at Course 1/Week 25: number analyzed (Participants) | 32 | 10 | 19 | 11 | 19
  Change at Course 1/Week 25 | -73.5 (28.74) | -74.1 (16.33) | -74.8 (25.21) | -59.9 (52.34) | -67.2 (28.49)
  Change at Course 2/Week 1 | -57.8 (80.94) | -51.0 (54.16) | -51.5 (46.11) | -60.8 (38.80) | -56.2 (45.29)
  Change at Course 2/Week 6: number analyzed (Participants) | 48 | 30 | 29 | 27 | 29
  Change at Course 2/Week 6 | -81.5 (26.08) | -64.6 (51.49) | -82.3 (21.43) | -73.2 (32.90) | -82.0 (20.56)
  Change at Course 2/Week 13: number analyzed (Participants) | 48 | 30 | 30 | 26 | 29
  Change at Course 2/Week 13 | -76.4 (31.23) | -54.7 (91.62) | -75.0 (34.02) | -76.8 (30.73) | -81.3 (26.43)
  Change at Course 2/Week 25: number analyzed (Participants) | 26 | 9 | 20 | 14 | 16
  Change at Course 2/Week 25 | -78.1 (24.72) | -84.4 (16.09) | -77.9 (21.66) | -76.1 (29.01) | -80.0 (21.86)
  Change at Course 3/Week 1 | -66.3 (55.96) | -59.9 (45.11) | -63.9 (39.07) | -74.3 (29.11) | -66.2 (31.33)
  Change at Course 3/Week 13: number analyzed (Participants) | 46 | 30 | 29 | 26 | 29
  Change at Course 3/Week 13 | -78.6 (36.94) | -70.4 (37.09) | -76.7 (29.14) | -84.0 (24.36) | -83.2 (26.99)
  Change at Course 3/Week 25: number analyzed (Participants) | 47 | 30 | 29 | 27 | 29
  Change at Course 3/Week 25 | -72.2 (46.88) | -51.5 (94.79) | -75.7 (29.79) | -79.1 (27.77) | -76.6 (37.50)

38. Primary Outcome: Percent Change From Initial Study Baseline in Individual Components of the ACR Response: Patient's Assessment of Arthritis Pain - by the End of Course 1
Description: Participants assessed the severity of their arthritis pain using a 100 millimeter (mm) VAS by placing a mark on the scale between 0 (no pain) and 100 (most severe pain), which corresponded to the magnitude of their pain.
Time Frame: Week 1, 6, 13, and 25 (Course 1).
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Percent change in score
Arm/Group | PF-05280586: by the End of Course 1 | Rituximab-EU: by the End of Course 1 | PF-05280586 (EU): by the End of Course 1 | Rituximab-US: by the End of Course 1 | PF-05280586 (US): by the End of Course 1
Number analyzed (Participants) | 58 | 32 | 33 | 30 | 30
Percent change in score
  Change at Course 1/Week 1 | -18.2 (67.42) | -36.3 (44.85) | -44.0 (58.90) | -38.8 (39.70) | -39.8 (27.60)
  Change at Course 1/Week 6: number analyzed (Participants) | 57 | 31 | 33 | 30 | 30
  Change at Course 1/Week 6 | -31.9 (79.38) | -51.5 (44.45) | -59.7 (33.09) | -42.5 (46.78) | -55.2 (28.28)
  Change at Course 1/Week 13: number analyzed (Participants) | 56 | 31 | 33 | 30 | 29
  Change at Course 1/Week 13 | -34.6 (52.28) | -42.4 (57.97) | -65.3 (28.79) | -54.8 (41.14) | -50.1 (30.48)
  Change at Course 1/Week 25: number analyzed (Participants) | 35 | 10 | 22 | 13 | 19
  Change at Course 1/Week 25 | -49.7 (35.41) | -19.6 (75.23) | -52.5 (42.73) | -32.7 (67.30) | -45.4 (32.50)

39. Primary Outcome: Percent Change From Initial Study Baseline in Individual Components of the ACR Response: Patient's Assessment of Arthritis Pain - by the End of Course 2
Description: as for outcome 38
Time Frame: Week 1, 6, 13, and 25 (Course 1 and Course 2).
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Percent change in score
Arm/Group | PF-05280586: by the End of Course 2 | Rituximab-EU/PF-05280586: by the End of Course 2 | PF-05280586 (EU): by the End of Course 2 | Rituximab-US/PF-05280586: by the End of Course 2 | PF-05280586 (US): by the End of Course 2
Number analyzed (Participants) | 54 | 30 | 31 | 29 | 29
Percent change in score
  Change at Course 1/Week 1 | -19.4 (68.24) | -34.9 (44.82) | -43.2 (59.94) | -37.1 (39.36) | -40.1 (28.05)
  Change at Course 1/Week 6 | -33.2 (80.43) | -50.1 (44.48) | -59.1 (33.46) | -40.9 (46.73) | -56.1 (28.28)
  Change at Course 1/Week 13 | -36.1 (51.66) | -40.5 (58.05) | -64.8 (29.18) | -53.4 (41.20) | -50.1 (30.48)
  Change at Course 1/Week 25: number analyzed (Participants) | 35 | 10 | 20 | 12 | 19
  Change at Course 1/Week 25 | -49.7 (35.41) | -19.6 (75.23) | -50.5 (43.76) | -31.0 (70.03) | -45.4 (32.50)
  Change at Course 2/Week 1 | -26.1 (77.23) | -36.4 (57.62) | -43.9 (46.93) | -40.6 (47.26) | -41.6 (30.62)
  Change at Course 2/Week 6: number analyzed (Participants) | 53 | 30 | 29 | 29 | 29
  Change at Course 2/Week 6 | -42.8 (69.12) | -50.5 (48.60) | -55.3 (30.66) | -60.1 (33.26) | -58.1 (26.39)
  Change at Course 2/Week 13: number analyzed (Participants) | 53 | 30 | 30 | 29 | 29
  Change at Course 2/Week 13 | -33.1 (61.98) | -40.6 (65.18) | -53.0 (42.09) | -36.0 (94.22) | -55.9 (28.76)
  Change at Course 2/Week 25: number analyzed (Participants) | 29 | 9 | 20 | 15 | 16
  Change at Course 2/Week 25 | -50.7 (41.77) | -59.4 (29.28) | -55.8 (31.08) | -44.8 (25.66) | -61.3 (24.95)

40. Primary Outcome: Percent Change From Initial Study Baseline in Individual Components of the ACR Response: Patient's Assessment of Arthritis Pain - by the End of Course 3
Description: as for outcome 38
Time Frame: Week 1, 6, 13, and 25 (Course 1 and Course 2), and Week 1, 13, and 25 (Course 3).
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Percent change in score
Arm/Group | PF-05280586: by the End of Course 3 | Rituximab-EU/PF-05280586/PF-05280586: by the End of Course 3 | PF-05280586 (EU): by the End of Course 3 | Rituximab-US/PF-05280586/PF-05280586: by the End of Course 3 | PF-05280586 (US): by the End of Course 3
Number analyzed (Participants) | 48 | 30 | 30 | 27 | 29
Percent change in score
  Change at Course 1/Week 1 | -19.1 (70.91) | -34.9 (44.82) | -41.6 (60.23) | -38.2 (40.64) | -40.1 (28.05)
  Change at Course 1/Week 6 | -31.8 (84.65) | -50.1 (44.48) | -58.0 (33.47) | -40.7 (48.45) | -56.1 (28.28)
  Change at Course 1/Week 13 | -39.2 (51.83) | -40.5 (58.05) | -63.8 (29.15) | -52.5 (42.60) | -50.1 (30.48)
  Change at Course 1/Week 25: number analyzed (Participants) | 32 | 10 | 19 | 11 | 19
  Change at Course 1/Week 25 | -49.0 (36.46) | -19.6 (75.23) | -48.4 (43.85) | -31.7 (73.41) | -45.4 (32.50)
  Change at Course 2/Week 1 | -26.4 (80.49) | -36.4 (57.62) | -42.5 (47.03) | -40.0 (48.91) | -41.6 (30.62)
  Change at Course 2/Week 6: number analyzed (Participants) | 48 | 30 | 29 | 27 | 29
  Change at Course 2/Week 6 | -41.1 (71.99) | -50.5 (48.60) | -55.3 (30.66) | -60.3 (34.45) | -58.1 (26.39)
  Change at Course 2/Week 13 | -33.9 (62.57) | -40.6 (65.18) | -53.0 (42.09) | -35.8 (97.72) | -55.9 (28.76)
  Change at Course 2/Week 25: number analyzed (Participants) | 26 | 9 | 20 | 14 | 16
  Change at Course 2/Week 25 | -56.7 (33.85) | -59.4 (29.28) | -55.8 (31.08) | -47.8 (23.72) | -61.3 (24.95)
  Change at Course 3/Week 1 | -24.0 (74.65) | -39.4 (50.56) | -37.2 (62.77) | -39.3 (44.07) | -45.3 (34.84)
  Change at Course 3/Week 13: number analyzed (Participants) | 46 | 30 | 29 | 26 | 29
  Change at Course 3/Week 13 | -37.9 (63.45) | -45.7 (52.35) | -57.9 (33.80) | -43.3 (50.22) | -55.7 (31.01)
  Change at Course 3/Week 25: number analyzed (Participants) | 47 | 30 | 30 | 27 | 29
  Change at Course 3/Week 25 | -28.5 (69.63) | -44.1 (45.48) | -53.9 (36.80) | -43.4 (62.71) | -53.9 (35.77)

41. Primary Outcome: Percent Change From Initial Study Baseline in Individual Components of the ACR Response: Patient's Global Assessment of Arthritis - by the End of Course 1
Description: Participants were asked the following question, "Considering all the ways your arthritis affects you, how are you feeling today?" Their response was recorded using a 100 mm VAS between 0 (very well) and 100 (very poor).
Time Frame: Week 1, 6, 13, and 25 (Course 1).
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Percent change in score
Arm/Group | PF-05280586: by the End of Course 1 | Rituximab-EU: by the End of Course 1 | PF-05280586 (EU): by the End of Course 1 | Rituximab-US: by the End of Course 1 | PF-05280586 (US): by the End of Course 1
Number analyzed (Participants) | 58 | 32 | 33 | 30 | 30
Percent change in score
  Change at Course 1/Week 1: number analyzed (Participants) | 57 | 32 | 33 | 30 | 29
  Change at Course 1/Week 1 | -18.9 (62.81) | -43.8 (41.27) | -40.3 (55.42) | -45.1 (32.92) | -39.2 (23.89)
  Change at Course 1/Week 6: number analyzed (Participants) | 57 | 31 | 33 | 30 | 30
  Change at Course 1/Week 6 | -34.6 (65.37) | -56.2 (34.62) | -56.8 (34.01) | -51.0 (33.61) | -58.3 (24.77)
  Change at Course 1/Week 13: number analyzed (Participants) | 55 | 31 | 33 | 30 | 29
  Change at Course 1/Week 13 | -39.1 (48.65) | -55.9 (46.04) | -62.0 (29.52) | -61.3 (29.78) | -56.2 (27.35)
  Change at Course 1/Week 25: number analyzed (Participants) | 35 | 10 | 22 | 13 | 19
  Change at Course 1/Week 25 | -52.6 (33.84) | -42.3 (52.55) | -48.4 (42.71) | -47.7 (22.70) | -46.5 (31.47)

42. Primary Outcome: Percent Change From Initial Study Baseline in Individual Components of the ACR Response: Patient's Global Assessment of Arthritis - by the End of Course 2
Description: as for outcome 41
Time Frame: Week 1, 6, 13, and 25 (Course 1 and Course 2).
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Percent change in score
Arm/Group | PF-05280586: by the End of Course 2 | Rituximab-EU/PF-05280586: by the End of Course 2 | PF-05280586 (EU): by the End of Course 2 | Rituximab-US/PF-05280586: by the End of Course 2 | PF-05280586 (US): by the End of Course 2
Number analyzed (Participants) | 54 | 30 | 31 | 29 | 29
Percent change in score
  Change at Course 1/Week 1: number analyzed (Participants) | 54 | 30 | 31 | 29 | 28
  Change at Course 1/Week 1 | -21.5 (62.57) | -41.7 (41.50) | -40.5 (55.52) | -43.8 (32.81) | -39.9 (24.05)
  Change at Course 1/Week 6 | -37.4 (64.66) | -55.0 (34.56) | -56.4 (34.31) | -49.7 (33.52) | -59.5 (24.29)
  Change at Course 1/Week 13 | -41.2 (47.09) | -54.6 (46.26) | -62.2 (29.35) | -60.3 (29.79) | -56.2 (27.35)
  Change at Course 1/Week 25: number analyzed (Participants) | 35 | 10 | 20 | 12 | 19
  Change at Course 1/Week 25 | -52.6 (33.84) | -42.3 (52.55) | -47.1 (43.42) | -46.3 (23.14) | -46.5 (31.47)
  Change at Course 2/Week 1 | -32.1 (62.08) | -41.9 (54.71) | -39.1 (45.93) | -50.6 (31.39) | -43.3 (27.34)
  Change at Course 2/Week 6: number analyzed (Participants) | 53 | 30 | 29 | 29 | 29
  Change at Course 2/Week 6 | -46.8 (46.61) | -51.5 (49.96) | -46.2 (49.97) | -62.0 (29.11) | -59.0 (25.26)
  Change at Course 2/Week 13: number analyzed (Participants) | 53 | 30 | 30 | 29 | 29
  Change at Course 2/Week 13 | -43.7 (40.69) | -45.1 (55.55) | -29.8 (142.51) | -53.3 (41.09) | -57.2 (23.56)
  Change at Course 2/Week 25: number analyzed (Participants) | 29 | 9 | 20 | 15 | 16
  Change at Course 2/Week 25 | -55.6 (33.12) | -59.1 (29.99) | -51.0 (33.35) | -47.3 (28.57) | -60.9 (21.76)

43. Primary Outcome: Percent Change From Initial Study Baseline in Individual Components of the ACR Response: Patient's Global Assessment of Arthritis - by the End of Course 3
Description: as for outcome 41
Time Frame: Week 1, 6, 13, and 25 (Course 1 and Course 2), and Week 1, 13, and 25 (Course 3).
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Percent change in score
Arm/Group | PF-05280586: by the End of Course 3 | Rituximab-EU/PF-05280586/PF-05280586: by the End of Course 3 | PF-05280586 (EU): by the End of Course 3 | Rituximab-US/PF-05280586/PF-05280586: by the End of Course 3 | PF-05280586 (US): by the End of Course 3
Number analyzed (Participants) | 48 | 30 | 30 | 27 | 29
Percent change in score
  Change at Course 1/Week 1: number analyzed (Participants) | 48 | 30 | 30 | 27 | 28
  Change at Course 1/Week 1 | -21.7 (65.60) | -41.7 (41.50) | -38.8 (55.71) | -44.4 (33.89) | -39.9 (24.05)
  Change at Course 1/Week 6 | -36.9 (67.42) | -55.0 (34.56) | -55.5 (34.55) | -50.2 (34.42) | -59.5 (24.29)
  Change at Course 1/Week 13 | -44.1 (48.95) | -54.6 (46.26) | -61.3 (29.42) | -60.1 (30.80) | -56.2 (27.35)
  Change at Course 1/Week 25: number analyzed (Participants) | 32 | 10 | 19 | 11 | 19
  Change at Course 1/Week 25 | -51.5 (35.06) | -42.3 (52.55) | -44.8 (43.28) | -47.4 (23.93) | -46.5 (31.47)
  Change at Course 2/Week 1 | -31.0 (65.11) | -41.9 (54.71) | -37.5 (45.85) | -50.2 (32.39) | -43.3 (27.34)
  Change at Course 2/Week 6: number analyzed (Participants) | 48 | 30 | 29 | 27 | 29
  Change at Course 2/Week 6 | -45.1 (48.34) | -51.5 (49.96) | -46.2 (49.97) | -63.5 (29.54) | -59.0 (25.26)
  Change at Course 2/Week 13 | -43.3 (41.50) | -45.1 (55.55) | -29.8 (142.51) | -54.7 (42.05) | -57.2 (23.56)
  Change at Course 2/Week 25: number analyzed (Participants) | 26 | 9 | 20 | 14 | 16
  Change at Course 2/Week 25 | -59.1 (31.65) | -59.1 (29.99) | -51.0 (33.35) | -49.9 (27.77) | -60.9 (21.76)
  Change at Course 3/Week 1 | -26.9 (63.81) | -45.4 (41.98) | -39.1 (46.90) | -42.9 (43.85) | -48.6 (34.18)
  Change at Course 3/Week 13: number analyzed (Participants) | 46 | 30 | 29 | 26 | 29
  Change at Course 3/Week 13 | -40.5 (48.27) | -52.6 (45.33) | -53.2 (34.27) | -52.3 (35.92) | -55.2 (28.16)
  Change at Course 3/Week 25: number analyzed (Participants) | 47 | 30 | 30 | 27 | 29
  Change at Course 3/Week 25 | -34.7 (50.49) | -43.3 (44.82) | -50.6 (39.52) | -53.9 (42.61) | -50.3 (44.57)

44. Primary Outcome: Percent Change From Initial Study Baseline in Individual Components of the ACR Response: Physician's Global Assessment of Arthritis - by the End of Course 1
Description: The investigator assessed how the participant's overall arthritis appeared at the time of the visit. This evaluation was based on the participant's disease signs, functional capacity and physical examination, and was independent of the Patient's Global Assessment of Arthritis. The investigator's response was recorded using a 100 mm VAS by placing a mark on the scale between 0 (very good) and 100 (very poor).
Time Frame: Week 1, 6, 13, and 25 (Course 1).
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Percent change in score
Arm/Group | PF-05280586: by the End of Course 1 | Rituximab-EU: by the End of Course 1 | PF-05280586 (EU): by the End of Course 1 | Rituximab-US: by the End of Course 1 | PF-05280586 (US): by the End of Course 1
Number analyzed (Participants) | 58 | 32 | 33 | 30 | 30
Percent change in score
  Change at Course 1/Week 1 | -40.3 (42.01) | -46.1 (42.81) | -54.2 (34.06) | -55.0 (26.03) | -52.4 (26.51)
  Change at Course 1/Week 6: number analyzed (Participants) | 57 | 31 | 33 | 30 | 30
  Change at Course 1/Week 6 | -60.4 (45.47) | -66.1 (40.40) | -71.3 (24.62) | -59.5 (39.66) | -73.0 (22.41)
  Change at Course 1/Week 13: number analyzed (Participants) | 56 | 31 | 33 | 30 | 29
  Change at Course 1/Week 13 | -69.3 (30.36) | -68.1 (37.74) | -76.1 (14.01) | -71.0 (27.86) | -69.9 (21.09)
  Change at Course 1/Week 25: number analyzed (Participants) | 35 | 10 | 22 | 13 | 19
  Change at Course 1/Week 25 | -67.0 (29.61) | -73.2 (25.00) | -71.4 (23.32) | -55.1 (28.56) | -59.9 (25.95)

45. Primary Outcome: Percent Change From Initial Study Baseline in Individual Components of the ACR Response: Physician's Global Assessment of Arthritis - by the End of Course 2
Description: as for outcome 44
Time Frame: Week 1, 6, 13, and 25 (Course 1 and Course 2).
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Percent change in score
Arm/Group | PF-05280586: by the End of Course 2 | Rituximab-EU/PF-05280586: by the End of Course 2 | PF-05280586 (EU): by the End of Course 2 | Rituximab-US/PF-05280586: by the End of Course 2 | PF-05280586 (US): by the End of Course 2
Number analyzed (Participants) | 54 | 30 | 31 | 29 | 29
Percent change in score
  Change at Course 1/Week 1 | -41.3 (42.20) | -45.4 (43.77) | -54.4 (33.27) | -54.0 (25.84) | -53.9 (25.58)
  Change at Course 1/Week 6 | -62.1 (44.83) | -65.1 (40.66) | -72.3 (23.31) | -58.5 (40.01) | -74.4 (21.44)
  Change at Course 1/Week 13 | -70.3 (28.43) | -67.2 (38.04) | -76.5 (13.39) | -70.3 (28.11) | -69.9 (21.09)
  Change at Course 1/Week 25: number analyzed (Participants) | 35 | 10 | 20 | 12 | 19
  Change at Course 1/Week 25 | -67.0 (29.61) | -73.2 (25.00) | -71.5 (22.98) | -54.7 (29.79) | -59.9 (25.95)
  Change at Course 2/Week 1: number analyzed (Participants) | 54 | 30 | 31 | 28 | 29
  Change at Course 2/Week 1 | -56.9 (50.62) | -49.5 (43.91) | -59.3 (28.59) | -56.6 (31.54) | -60.7 (23.54)
  Change at Course 2/Week 6: number analyzed (Participants) | 53 | 30 | 29 | 29 | 29
  Change at Course 2/Week 6 | -76.4 (26.53) | -66.9 (36.14) | -74.0 (24.77) | -69.4 (25.81) | -74.6 (21.81)
  Change at Course 2/Week 13: number analyzed (Participants) | 53 | 30 | 30 | 29 | 29
  Change at Course 2/Week 13 | -74.0 (24.66) | -64.6 (44.61) | -72.1 (22.92) | -69.0 (35.02) | -72.9 (30.55)
  Change at Course 2/Week 25: number analyzed (Participants) | 29 | 9 | 20 | 15 | 16
  Change at Course 2/Week 25 | -68.5 (26.40) | -73.7 (21.26) | -71.9 (27.15) | -58.9 (34.65) | -68.7 (32.49)

46. Primary Outcome: Percent Change From Initial Study Baseline in Individual Components of the ACR Response: Physician's Global Assessment of Arthritis - by the End of Course 3
Description: as for outcome 44
Time Frame: Week 1, 6, 13, and 25 (Course 1 and Course 2), and Week 1, 13, and 25 (Course 3).
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Percent change in score
Arm/Group | PF-05280586: by the End of Course 3 | Rituximab-EU/PF-05280586/PF-05280586: by the End of Course 3 | PF-05280586 (EU): by the End of Course 3 | Rituximab-US/PF-05280586/PF-05280586: by the End of Course 3 | PF-05280586 (US): by the End of Course 3
Number analyzed (Participants) | 48 | 30 | 30 | 27 | 29
Percent change in score
  Change at Course 1/Week 1 | -39.7 (43.82) | -45.4 (43.77) | -53.1 (32.94) | -55.6 (25.07) | -53.9 (25.58)
  Change at Course 1/Week 6 | -62.8 (45.89) | -65.1 (40.66) | -71.6 (23.44) | -61.0 (40.38) | -74.4 (21.44)
  Change at Course 1/Week 13 | -72.5 (29.26) | -67.2 (38.04) | -76.0 (13.34) | -70.5 (29.13) | -69.9 (21.09)
  Change at Course 1/Week 25: number analyzed (Participants) | 32 | 10 | 19 | 11 | 19
  Change at Course 1/Week 25 | -65.9 (30.76) | -73.2 (25.00) | -70.4 (22.98) | -60.1 (24.56) | -59.9 (25.95)
  Change at Course 2/Week 1: number analyzed (Participants) | 48 | 30 | 30 | 26 | 29
  Change at Course 2/Week 1 | -57.2 (53.03) | -49.5 (43.91) | -58.2 (28.45) | -56.2 (31.66) | -60.7 (23.54)
  Change at Course 2/Week 6: number analyzed (Participants) | 48 | 30 | 29 | 27 | 29
  Change at Course 2/Week 6 | -75.3 (27.47) | -66.9 (36.14) | -74.0 (24.77) | -70.2 (26.55) | -74.6 (21.81)
  Change at Course 2/Week 13 | -73.4 (25.64) | -64.6 (44.61) | -72.1 (22.92) | -69.7 (36.19) | -72.9 (30.55)
  Change at Course 2/Week 25: number analyzed (Participants) | 26 | 9 | 20 | 14 | 16
  Change at Course 2/Week 25 | -70.6 (24.17) | -73.7 (21.26) | -71.9 (27.15) | -63.8 (30.10) | -68.7 (32.49)
  Change at Course 3/Week 1 | -52.6 (55.21) | -54.6 (43.47) | -59.6 (29.85) | -52.8 (44.20) | -62.9 (28.65)
  Change at Course 3/Week 13: number analyzed (Participants) | 46 | 30 | 29 | 26 | 28
  Change at Course 3/Week 13 | -74.6 (33.44) | -62.3 (54.14) | -73.3 (19.12) | -71.5 (22.57) | -73.0 (23.11)
  Change at Course 3/Week 25: number analyzed (Participants) | 47 | 30 | 28 | 27 | 29
  Change at Course 3/Week 25 | -74.0 (25.59) | -59.9 (42.55) | -74.3 (20.48) | -72.7 (23.30) | -70.9 (26.63)

47. Primary Outcome: Percent Change From Initial Study Baseline in Individual Components of the ACR Response: Health Assessment Questionnaire - Disability Index (HAQ-DI) - by the End of Course 1
Description: HAQ-DI assessed the degree of difficulty participants experienced in 8 daily living activity domains during a week: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and other activities. Each activity category consisted of 2-3 items. Each question's difficulty was scored from 0-3 (0=no difficulty, 1=some difficulty, 2=much difficulty, 3=unable to do). Activities requiring assistance (from people or assistive devices) were adjusted to ≥2 to denote more limited functional status. The questionnaire was to be completed by the participant prior to any procedures during the visit, if possible.
  Overall HAQ-DI score was computed as the sum of domain scores divided by the number of domains answered, providing a score from 0-3. Low scores denoted improvement of disability/lower degree of domain difficulty.
  Primary outcomes reported post baseline mean percent (%) changes in HAQ-DI score. Post baseline values are reported on the % change from initial study Baseline scale.
Time Frame: Week 1, 6, 13, and 25 (Course 1).
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Percent change in score
Arm/Group | PF-05280586: by the End of Course 1 | Rituximab-EU: by the End of Course 1 | PF-05280586 (EU): by the End of Course 1 | Rituximab-US: by the End of Course 1 | PF-05280586 (US): by the End of Course 1
Number analyzed (Participants) | 58 | 32 | 33 | 30 | 30
Percent change in score
  Change at Course 1/Week 1 | -12.2 (54.91) | -31.0 (38.52) | -39.1 (45.85) | -28.8 (33.42) | -27.7 (36.15)
  Change at Course 1/Week 6: number analyzed (Participants) | 57 | 31 | 33 | 30 | 30
  Change at Course 1/Week 6 | -20.0 (48.09) | -39.1 (38.66) | -45.8 (35.63) | -35.9 (30.65) | -31.7 (36.38)
  Change at Course 1/Week 13: number analyzed (Participants) | 56 | 31 | 33 | 30 | 29
  Change at Course 1/Week 13 | -17.7 (41.95) | -40.0 (43.21) | -47.5 (34.34) | -30.0 (37.25) | -35.8 (33.09)
  Change at Course 1/Week 25: number analyzed (Participants) | 35 | 10 | 22 | 13 | 19
  Change at Course 1/Week 25 | -26.3 (42.52) | -24.1 (32.50) | -43.6 (38.36) | -33.9 (39.17) | -27.2 (41.12)

48. Primary Outcome: Percent Change From Initial Study Baseline in Individual Components of the ACR Response: Health Assessment Questionnaire - Disability Index (HAQ-DI) - by the End of Course 2
Description: as for outcome 47
Time Frame: Week 1, 6, 13, and 25 (Course 1 and Course 2).
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Percent change in score
Arm/Group | PF-05280586: by the End of Course 2 | Rituximab-EU/PF-05280586: by the End of Course 2 | PF-05280586 (EU): by the End of Course 2 | Rituximab-US/PF-05280586: by the End of Course 2 | PF-05280586 (US): by the End of Course 2
Number analyzed (Participants) | 54 | 30 | 31 | 29 | 29
Percent change in score
  Change at Course 1/Week 1 | -15.6 (45.37) | -29.3 (37.54) | -40.0 (43.05) | -26.7 (32.08) | -28.4 (36.53)
  Change at Course 1/Week 6 | -23.4 (41.60) | -37.1 (37.61) | -46.8 (31.78) | -34.1 (29.58) | -32.6 (36.66)
  Change at Course 1/Week 13 | -21.6 (34.03) | -38.0 (42.46) | -48.4 (31.07) | -28.0 (36.26) | -35.8 (33.09)
  Change at Course 1/Week 25: number analyzed (Participants) | 35 | 10 | 20 | 12 | 19
  Change at Course 1/Week 25 | -26.3 (42.52) | -24.1 (32.50) | -44.0 (35.30) | -31.5 (39.92) | -27.2 (41.12)
  Change at Course 2/Week 1 | -19.4 (44.16) | -36.6 (41.08) | -44.9 (34.41) | -24.2 (35.47) | -27.6 (32.91)
  Change at Course 2/Week 6: number analyzed (Participants) | 53 | 30 | 29 | 29 | 29
  Change at Course 2/Week 6 | -27.3 (42.86) | -38.2 (41.14) | -44.1 (38.55) | -27.2 (40.71) | -35.4 (44.10)
  Change at Course 2/Week 13: number analyzed (Participants) | 53 | 30 | 30 | 29 | 29
  Change at Course 2/Week 13 | -24.9 (44.40) | -38.5 (40.36) | -45.3 (41.12) | -28.4 (38.05) | -32.3 (64.88)
  Change at Course 2/Week 25: number analyzed (Participants) | 29 | 9 | 20 | 15 | 16
  Change at Course 2/Week 25 | -23.4 (79.52) | -30.7 (37.00) | -43.2 (38.79) | -22.3 (29.32) | -48.7 (27.77)

49. Primary Outcome: Percent Change From Initial Study Baseline in Individual Components of the ACR Response: Health Assessment Questionnaire - Disability Index (HAQ-DI) - by the End of Course 3
Description: as for outcome 47
Time Frame: Week 1, 6, 13, and 25 (Course 1 and Course 2), and Week 1, 13, and 25 (Course 3).
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Percent change in score
Arm/Group | PF-05280586: by the End of Course 3 | Rituximab-EU/PF-05280586/PF-05280586: by the End of Course 3 | PF-05280586 (EU): by the End of Course 3 | Rituximab-US/PF-05280586/PF-05280586: by the End of Course 3 | PF-05280586 (US): by the End of Course 3
Number analyzed (Participants) | 48 | 30 | 30 | 27 | 29
Percent change in score
  Change at Course 1/Week 1 | -13.9 (46.19) | -29.3 (37.54) | -38.6 (42.99) | -26.7 (31.76) | -28.4 (36.53)
  Change at Course 1/Week 6 | -23.1 (42.48) | -37.1 (37.61) | -45.2 (31.03) | -33.4 (30.08) | -32.6 (36.66)
  Change at Course 1/Week 13 | -23.2 (35.62) | -38.0 (42.46) | -46.8 (30.36) | -27.7 (37.07) | -35.8 (33.09)
  Change at Course 1/Week 25: number analyzed (Participants) | 32 | 10 | 19 | 11 | 19
  Change at Course 1/Week 25 | -26.7 (44.36) | -24.1 (32.50) | -41.3 (34.12) | -30.2 (41.61) | -27.2 (41.12)
  Change at Course 2/Week 1 | -18.8 (45.07) | -36.6 (41.08) | -43.2 (33.71) | -24.3 (36.60) | -27.6 (32.91)
  Change at Course 2/Week 6: number analyzed (Participants) | 48 | 30 | 29 | 27 | 29
  Change at Course 2/Week 6 | -26.6 (43.60) | -38.2 (41.14) | -44.1 (38.55) | -26.6 (42.19) | -35.4 (44.10)
  Change at Course 2/Week 13 | -22.9 (44.48) | -38.5 (40.36) | -45.3 (41.12) | -27.2 (39.12) | -32.3 (64.88)
  Change at Course 2/Week 25: number analyzed (Participants) | 26 | 9 | 20 | 14 | 16
  Change at Course 2/Week 25 | -21.0 (82.68) | -30.7 (37.00) | -43.2 (38.79) | -25.0 (28.30) | -48.7 (27.77)
  Change at Course 3/Week 1 | -18.7 (54.57) | -37.2 (41.42) | -41.5 (47.06) | -20.4 (43.26) | -22.5 (60.13)
  Change at Course 3/Week 13: number analyzed (Participants) | 46 | 30 | 29 | 26 | 29
  Change at Course 3/Week 13 | -25.3 (43.76) | -32.6 (42.25) | -40.8 (50.01) | -24.8 (36.50) | -40.7 (44.12)
  Change at Course 3/Week 25: number analyzed (Participants) | 47 | 30 | 30 | 27 | 29
  Change at Course 3/Week 25 | -23.7 (42.05) | -37.7 (42.58) | -48.7 (29.85) | -31.1 (32.38) | -34.5 (46.20)

50. Primary Outcome: Outcome Measure Using HAQ-DI - by the End of Course 1
Description: HAQ-DI assessed the degree of difficulty participants experienced in 8 daily living activity domains during a week: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and other activities. Each activity category consisted of 2-3 items. Each question's difficulty was scored from 0-3 (0=no difficulty, 1=some difficulty, 2=much difficulty, 3=unable to do). Activities requiring assistance (from people or assistive devices) were adjusted to ≥2 to denote more limited functional status. The questionnaire was to be completed by the participant prior to any procedures during the visit, if possible.
  Overall HAQ-DI score was computed as the sum of domain scores divided by the number of domains answered, providing a score from 0-3. Low scores denoted improvement of disability/lower degree of domain difficulty.
  Primary outcome reported in the table is mean HAQ-DI score at each time point, and it is on the scale of HAQ-DI score with the range from 0 to 3.
Time Frame: Week 1, 6, 13, and 25 (Course 1).
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | PF-05280586: by the End of Course 1 | Rituximab-EU: by the End of Course 1 | PF-05280586 (EU): by the End of Course 1 | Rituximab-US: by the End of Course 1 | PF-05280586 (US): by the End of Course 1
Number analyzed (Participants) | 58 | 32 | 33 | 30 | 30
Score on a scale
  Course 1/Week 1 | 1.4 (0.66) | 1.1 (0.73) | 1.0 (0.63) | 1.2 (0.71) | 1.3 (0.78)
  Course 1/Week 6: number analyzed (Participants) | 57 | 31 | 33 | 30 | 30
  Course 1/Week 6 | 1.3 (0.70) | 1.0 (0.68) | 0.9 (0.62) | 1.1 (0.66) | 1.2 (0.75)
  Course 1/Week 13: number analyzed (Participants) | 56 | 31 | 33 | 30 | 29
  Course 1/Week 13 | 1.3 (0.63) | 1.0 (0.74) | 0.8 (0.59) | 1.2 (0.65) | 1.1 (0.70)
  Course 1/Week 25: number analyzed (Participants) | 35 | 10 | 22 | 13 | 19
  Course 1/Week 25 | 1.2 (0.60) | 1.3 (0.67) | 0.9 (0.65) | 1.1 (0.75) | 1.1 (0.66)

51. Primary Outcome: Outcome Measure Using HAQ-DI - by the End of Course 2
Description: as for outcome 50
Time Frame: Week 1, 6, 13, and 25 (Course 1 and Course 2).
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | PF-05280586: by the End of Course 2 | Rituximab-EU/PF-05280586: by the End of Course 2 | PF-05280586 (EU): by the End of Course 2 | Rituximab-US/PF-05280586: by the End of Course 2 | PF-05280586 (US): by the End of Course 2
Number analyzed (Participants) | 54 | 30 | 31 | 29 | 29
Score on a scale
  Course 1/Week 1 | 1.4 (0.68) | 1.2 (0.72) | 1.0 (0.60) | 1.3 (0.70) | 1.2 (0.77)
  Course 1/Week 6 | 1.3 (0.71) | 1.0 (0.66) | 0.9 (0.60) | 1.1 (0.66) | 1.1 (0.73)
  Course 1/Week 13 | 1.3 (0.64) | 1.0 (0.73) | 0.8 (0.58) | 1.2 (0.64) | 1.1 (0.70)
  Course 1/Week 25: number analyzed (Participants) | 35 | 10 | 20 | 12 | 19
  Course 1/Week 25 | 1.2 (0.60) | 1.3 (0.67) | 0.9 (0.63) | 1.1 (0.78) | 1.1 (0.66)
  Course 2/Week 1 | 1.3 (0.66) | 1.0 (0.75) | 0.9 (0.64) | 1.3 (0.69) | 1.2 (0.75)
  Course 2/Week 6: number analyzed (Participants) | 53 | 30 | 29 | 29 | 29
  Course 2/Week 6 | 1.2 (0.67) | 1.0 (0.69) | 0.9 (0.60) | 1.2 (0.61) | 1.0 (0.65)
  Course 2/Week 13: number analyzed (Participants) | 53 | 30 | 30 | 29 | 29
  Course 2/Week 13 | 1.2 (0.69) | 1.0 (0.69) | 0.9 (0.60) | 1.2 (0.65) | 1.0 (0.67)
  Course 2/Week 25: number analyzed (Participants) | 29 | 9 | 20 | 15 | 16
  Course 2/Week 25 | 1.1 (0.71) | 1.2 (0.75) | 0.9 (0.69) | 1.4 (0.75) | 0.8 (0.60)

52. Primary Outcome: Outcome Measure Using HAQ-DI - by the End of Course 3
Description: as for outcome 50
Time Frame: Week 1, 6, 13, and 25 (Course 1 and Course 2), and Week 1, 13, and 25 (Course 3).
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | PF-05280586: by the End of Course 3 | Rituximab-EU/PF-05280586/PF-05280586: by the End of Course 3 | PF-05280586 (EU): by the End of Course 3 | Rituximab-US/PF-05280586/PF-05280586: by the End of Course 3 | PF-05280586 (US): by the End of Course 3
Number analyzed (Participants) | 48 | 30 | 30 | 27 | 29
Score on a scale
  Course 1/Week 1 | 1.4 (0.67) | 1.2 (0.72) | 1.0 (0.60) | 1.3 (0.70) | 1.2 (0.77)
  Course 1/Week 6 | 1.2 (0.69) | 1.0 (0.66) | 0.9 (0.60) | 1.2 (0.67) | 1.1 (0.73)
  Course 1/Week 13 | 1.2 (0.62) | 1.0 (0.73) | 0.9 (0.57) | 1.2 (0.65) | 1.1 (0.70)
  Course 1/Week 25: number analyzed (Participants) | 32 | 10 | 19 | 11 | 19
  Course 1/Week 25 | 1.1 (0.59) | 1.3 (0.67) | 1.0 (0.62) | 1.1 (0.80) | 1.1 (0.66)
  Course 2/Week 1 | 1.3 (0.64) | 1.0 (0.75) | 0.9 (0.64) | 1.3 (0.71) | 1.2 (0.75)
  Course 2/Week 6: number analyzed (Participants) | 48 | 30 | 29 | 27 | 29
  Course 2/Week 6 | 1.2 (0.66) | 1.0 (0.69) | 0.9 (0.60) | 1.2 (0.63) | 1.0 (0.65)
  Course 2/Week 13 | 1.2 (0.69) | 1.0 (0.69) | 0.9 (0.60) | 1.2 (0.66) | 1.0 (0.67)
  Course 2/Week 25: number analyzed (Participants) | 26 | 9 | 20 | 14 | 16
  Course 2/Week 25 | 1.1 (0.66) | 1.2 (0.75) | 0.9 (0.69) | 1.3 (0.77) | 0.8 (0.60)
  Course 3/Week 1 | 1.3 (0.67) | 1.0 (0.71) | 0.9 (0.64) | 1.3 (0.72) | 1.1 (0.71)
  Course 3/Week 13: number analyzed (Participants) | 46 | 30 | 29 | 26 | 29
  Course 3/Week 13 | 1.2 (0.67) | 1.1 (0.74) | 0.9 (0.54) | 1.2 (0.67) | 0.9 (0.66)
  Course 3/Week 25 (EOT): number analyzed (Participants) | 47 | 30 | 30 | 27 | 29
  Course 3/Week 25 (EOT) | 1.2 (0.68) | 1.0 (0.77) | 0.9 (0.60) | 1.2 (0.68) | 1.0 (0.71)

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) were logged from informed consent until up to 28 calendar days after last study drug administration or Long Term Follow-Up, whichever was last. Adverse events (AEs) were logged from first dose of study drug to last visit.
Description: SAEs & AEs were summarized by course for events with first onset on or after the first dose of study drug in that course & before the first dose of in the subsequent course, or any pre-existing event that worsened in severity during that course. An event may appear twice as data is cumulative for participants who received treatment in Course 2 & 3.
Arm/Group | PF-05280586: by the End of Course 1 | Rituximab-EU: by the End of Course 1 | PF-05280586 (EU): by the End of Course 1 | Rituximab-US: by the End of Course 1 | PF-05280586 (US): by the End of Course 1 | PF-05280586: by the End of Course 2 | Rituximab-EU/PF-05280586: by the End of Course 2 | PF-05280586 (EU): by the End of Course 2 | Rituximab-US/PF-05280586: by the End of Course 2 | PF-05280586 (US): by the End of Course 2 | PF-05280586: by the End of Course 3 | Rituximab-EU/PF-05280586/PF-05280586: by the End of Course 3 | PF-05280586 (EU): by the End of Course 3 | Rituximab-US/PF-05280586/PF-05280586: by the End of Course 3 | PF-05280586 (US): by the End of Course 3
Serious Adverse Events (participants affected / at risk) | 4/58 | 2/32 | 2/33 | 1/30 | 2/30 | 6/54 | 1/30 | 4/31 | 2/29 | 1/29 | 4/48 | 1/30 | 4/30 | 1/27 | 1/29
Other Adverse Events (participants affected / at risk) | 18/58 | 3/32 | 8/33 | 15/30 | 7/30 | 26/54 | 15/30 | 13/31 | 18/29 | 10/29 | 25/48 | 18/30 | 15/30 | 18/27 | 17/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-05280586: by the End of Course 1 (N=58) | Rituximab-EU: by the End of Course 1 (N=32) | PF-05280586 (EU): by the End of Course 1 (N=33) | Rituximab-US: by the End of Course 1 (N=30) | PF-05280586 (US): by the End of Course 1 (N=30) | PF-05280586: by the End of Course 2 (N=54) | Rituximab-EU/PF-05280586: by the End of Course 2 (N=30) | PF-05280586 (EU): by the End of Course 2 (N=31) | Rituximab-US/PF-05280586: by the End of Course 2 (N=29) | PF-05280586 (US): by the End of Course 2 (N=29) | PF-05280586: by the End of Course 3 (N=48) | Rituximab-EU/PF-05280586/PF-05280586: by the End of Course 3 (N=30) | PF-05280586 (EU): by the End of Course 3 (N=30) | Rituximab-US/PF-05280586/PF-05280586: by the End of Course 3 (N=27) | PF-05280586 (US): by the End of Course 3 (N=29)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pericarditis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diaphragmatic Hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Inguinal Hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Umbilical Hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Arthritis Infective (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastroenteritis Viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 2 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ureterolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Subcutaneous Abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wound Infection Staphylococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blighted Ovum (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Arthritis Bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Transient Ischemic Attack (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PF-05280586: by the End of Course 1 (N=58) | Rituximab-EU: by the End of Course 1 (N=32) | PF-05280586 (EU): by the End of Course 1 (N=33) | Rituximab-US: by the End of Course 1 (N=30) | PF-05280586 (US): by the End of Course 1 (N=30) | PF-05280586: by the End of Course 2 (N=54) | Rituximab-EU/PF-05280586: by the End of Course 2 (N=30) | PF-05280586 (EU): by the End of Course 2 (N=31) | Rituximab-US/PF-05280586: by the End of Course 2 (N=29) | PF-05280586 (US): by the End of Course 2 (N=29) | PF-05280586: by the End of Course 3 (N=48) | Rituximab-EU/PF-05280586/PF-05280586: by the End of Course 3 (N=30) | PF-05280586 (EU): by the End of Course 3 (N=30) | Rituximab-US/PF-05280586/PF-05280586: by the End of Course 3 (N=27) | PF-05280586 (US): by the End of Course 3 (N=29)
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1 | 2 | 2 | 2 | 1 | 1 | 3 | 2 | 1 | 1 | 1 | 3 | 2
Nausea (Gastrointestinal disorders) | 2 | 0 | 1 | 2 | 0 | 4 | 0 | 1 | 2 | 2 | 3 | 0 | 1 | 1 | 2
Vomiting (Gastrointestinal disorders) | 1 | 0 | 2 | 2 | 0 | 2 | 1 | 2 | 2 | 1 | 2 | 1 | 2 | 1 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 3 | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 3 | 1 | 1 | 1 | 1 | 4 | 1 | 3 | 2 | 2 | 4 | 1 | 4 | 3
Urinary Tract Infection (Infections and infestations) | 4 | 0 | 1 | 0 | 1 | 5 | 1 | 1 | 0 | 2 | 5 | 1 | 3 | 1 | 2
Foot Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 1 | 2 | 2 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 2 | 0 | 2 | 0 | 2 | 2 | 0 | 2 | 0 | 2 | 2 | 0
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 4 | 1 | 3 | 1 | 1 | 5 | 2 | 3 | 2 | 2 | 5 | 3 | 3 | 2 | 2
Dizziness (Nervous system disorders) | 1 | 0 | 1 | 2 | 0 | 2 | 0 | 1 | 2 | 1 | 2 | 1 | 1 | 1 | 1
Headache (Nervous system disorders) | 1 | 0 | 0 | 2 | 0 | 2 | 0 | 1 | 2 | 1 | 1 | 0 | 2 | 1 | 1
Depression (Psychiatric disorders) | 1 | 0 | 0 | 2 | 0 | 2 | 1 | 0 | 2 | 0 | 3 | 1 | 0 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 2 | 0 | 3 | 0 | 1 | 2 | 0 | 2 | 0 | 1 | 2 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 2
Skin Lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 2 | 0
Oedema Peripheral (General disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 0 | 1 | 2 | 1 | 3 | 0
Bronchitis (Infections and infestations) | 2 | 1 | 0 | 1 | 0 | 4 | 2 | 1 | 2 | 1 | 5 | 2 | 2 | 3 | 2
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 3 | 0 | 1 | 0 | 1 | 1 | 2
Oral Candidiasis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 1 | 1 | 1 | 1 | 1 | 4 | 2 | 2 | 2 | 2 | 4 | 2 | 2 | 2 | 2
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 1 | 1 | 0 | 1 | 3 | 2 | 1 | 0
Neutrophil Count Decreased (Investigations) | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0
Vitamin D Deficiency (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 1 | 2 | 1 | 0
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 2
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Gastrointestinal Viral Infection (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 1
Oral Herpes (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 1
Wrist Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 2
Alanine Aminotransferase Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 2
Aspartate Aminotransferase Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2
White Blood Cell Count Decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 60 days from the time submitted to the sponsor for review. The sponsor cannot extend the embargo. Investigator will, on request, remove any previously undisclosed Confidential Information (other than the Study results themselves) before disclosure.